

# STATISTICAL ANALYSIS PLAN

# FOR CLINICAL STUDY REPORT AC-065A309

# A MULTICENTER, OPEN-LABEL, SINGLE-SEQUENCE CROSS-OVER STUDY TO ASSESS SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF INTRAVENOUS SELEXIPAG IN SUBJECTS WITH STABLE PULMONARY ARTERIAL HYPERTENSION SWITCHING FROM AN ORAL STABLE DOSE OF SELEXIPAG

Purpose of Analysis Clinical Study Report

Investigational Drug Selexipag / ACT-293987

Protocol Number AC-065A309
Actelion Document Number D-18.239
Document Status/Version Number Final 2.0
Date 2 July 2018

Author CRO Trial Statistician

Reviewer Clinical Science Program Head /

Clinical Trial Physician

Reviewer Clinical Pharmacologist

Reviewer Medical Writer
Reviewer Medical Writer

Reviewer Clinical Trial Scientist

Reviewer Drug Safety Physician
Reviewer Senior Expert Statistician


Property of Actelion Pharmaceuticals Ltd. May not be used, divulged, published or otherwise disclosed without the consent of Actelion Pharmaceuticals Ltd.

# **TABLE OF CONTENTS**

| LI | ST OF ABBI | REVIATIONS AND ACRONYMS | 6 |
|---|---|---|---|
| 1 | INTRODU | CTION | 8 |
| 2 | STUDY DI | ESIGN AND FLOW | 8 |
| | 2.1 St | udy design | 8 |
| | | udy visit and assessment schedule | |
| | | nalysis periods | |
| | | andomization and blinding | |
| | | imple Size | |
| 3 | OBJECTIV | 'ES | 11 |
| | 3.1 Pr | imary objective | 11 |
| | | ther objectives | |
| 4 | ANALYSI | S SETS | 12 |
| | 4.1 De | efinitions of analysis sets | 12 |
| | 4.1.1 | Screened Analysis Set | |
| | 4.1.2 | Full Analysis Šet | |
| | 4.1.3 | Safety Analysis Set | 12 |
| | 4.1.4 | i.v. Safety Analysis Set | 12 |
| | 4.1.5 | Pharmacokinetic Analysis Set | 12 |
| | 4.2 Us | sage of the analysis sets | 14 |
| 5 | STUDY SU | JBJECTS VARIABLES AND ANALYSES | 15 |
| | 5.1 Su | ubject disposition | 15 |
| | 5.1.1 | Subject disposition and enrollment into analysis periods | |
| | 5.1.2 | Screening failures | |
| | 5.1.3 | Study completion/discontinuation | 15 |
| | 5.1.4 | Study treatment completion/discontinuation | 16 |
| | 5.2 Pr | otocol deviations | 16 |
| | 5.3 Ex | clusion from analysis sets | 16 |
| | 5.4 Su | ıbject characteristics | |
| | 5.4.1 | Demographics | |
| | 5.4.2 | Baseline disease characteristics | |
| | 5.4.3 | Other baseline characteristics | |
| | 5.4.4 | Medical history | |
| | 5.4.5 | Previous and concomitant therapies | |
| | 5.5 St | udy treatment exposure and compliance | 19 |

| | 5.5.1 | Exposure | 19 |
|---|---|---|---|
| | 5.5.2 | Compliance with study treatment | |
| 6 | EFFICACY | VARIABLES AND ANALYSES | 20 |
| 7 | SAFETY VA | ARIABLES | 20 |
| | 7.1 Ove | erview of safety analyses including subgroup analyses | 20 |
| | 7.1.1 | Overview of safety and tolerability endpoints | |
| | 7.2 Adv | /erse events | |
| | 7.2.1 | Variables | 22 |
| | 7.2.2 | Analysis | 24 |
| | 7.3 Dea | ıths | 26 |
| | 7.4 Lab | oratory | 26 |
| | 7.4.1 | Measurements | 26 |
| | 7.4.2 | Variables | 27 |
| | 7.4.3 | Analysis | 27 |
| | 7.5 Vita | al signs, physical findings, and other observations related to safety. | |
| | 7.5.1 | Vital signs | 28 |
| | 7.5.2 | Physical findings | 30 |
| | 7.5.3 | WHO functional class | 31 |
| | 7.6 Elec | ctrocardiograph | 31 |
| | 7.6.1 | Variables | 31 |
| | 7.6.2 | Variables | 32 |
| | 7.6.3 | Analysis | 33 |
| | 7.7 Sub | group analysis of safety variables | 34 |
| | 7.8 Pha | rmacokinetic variables | 34 |
| | 7.8.1 | Measurements | 34 |
| | 7.8.2 | Pharmacokinetic endpoints | 34 |
| | 7.8.3 | Pharmacokinetic variables | |
| | 7.8.4 | Analysis | 35 |
| 8 | GENERAL S | STATISTICAL METHODOLOGY | 37 |
| | 8.1 Gen | neral rules for data presentations | 37 |
| | 8.1.1 | Summary statistics of non-PK data | |
| | 8.1.2 | Summary statistics of PK data | |
| | 8.2 Stat | istical methods | |
| | 8.2.1 | Statistical methods for discrete data | |
| | 8.2.2 | Statistical methods for continuous data | |
| 9 | INTERIM A | NALYSIS | 41 |
| 10 | GENERAL I | DEFINITIONS AND DERIVATIONS | 41 |

# Confidential

| | 10.1 H | andling of screening and re-screening data | 41 |
|---|---|---|---|
| | 10.2 A | nalysis periods and visit windows | 41 |
| | 10.2.1 | | |
| | 10.2.2 | Study days | 41 |
| | 10.2.3 | | |
| | 10.2.4 | Unscheduled visits and visit windows | 41 |
| | 10.3 U | ptravi dosage subgroups | 42 |
| | 10.4 D | Perived and computed variables for analysis datasets | 42 |
| | 10.5 H | andling of missing/incomplete date and time fields | 42 |
| | 10.6 H | andling of missing infusion durations | 43 |
| 11 | | S OR CLARIFICATIONS TO ANALYSES PLANNED IN THE ROTOCOL | 43 |
| | 11.1 C | hanges to the analyses planned in the study protocol | 43 |
| | | hanges in the conduct of the study / data collection | |
| | 11.3 C | larifications concerning endpoint definitions and related variables or | |
| | S1 | atistical methods | 43 |
| | 11.3.1 | <b>1</b> | |
| | 11.3.2 | Additional analyses as compared to the study protocol | 44 |
| 12 | LIST OF T | TABLES, LISTINGS AND FIGURES | 44 |
| 13 | REFEREN | ICES | 57 |
| 1 / | A DDENIDI | CES | <b>5</b> 0 |

# LIST OF TABLES

| Table 1 | Study documents | 8 |
|---|---|---|
| Table 2 | Summary of analysis periods | 10 |
| Table 3 | Protocol deviations leading to an exclusion from the PKS | |
| | Γable 4 Overview of the different analysis sets and their usage | |
| Table 5 | PAH-specific therapies. | 18 |
| Table 6 | Correspondence of i.v. selexipag dose compared to Uptravi oral doses | 20 |
| Table 7 | Overview of safety and tolerability endpoints and populations in planned analysis periods | |
| Table 8 | Overview of adverse event analyses | |
| Table 9 | Schedule vital signs monitoring in Period 2 | |
| Table 10 | Marked abnormalities in blood pressure | |
| Table 11 | Pre-specified ECG findings categories | |
| Table 12 | QT prolongations in ECG parameters | |
| Table 13 | Analysis visit windows | |
| Table 14 Thresholds for marked laboratory abnormalities | | |
| Figure 1 | LIST OF FIGURES Study design and flow | 10 |
| | LIST OF APPENDICES | |
| Appendix A | Protocol synopsis | |
| Appendix B | Visit and assessment schedule | 63 |
| Appendix C | Discussion and further considerations of the applied statistical | |
| | methods | |
| Appendix D | Definitions of marked abnormalities and elevated liver function tests | |
| Appendix E | Mock layout | |
| Appendix F | Document history | 135 |

# LIST OF ABBREVIATIONS AND ACRONYMS

| AE | Adverse event |
|---|---|
| ADaM | Analysis data model |
| ALT | Alanine aminotransferase |
| AP | Alkaline phosphatase |
| AST | Aspartate aminotransferase |
| ATC | Anatomic Therapeutic Chemical |
| $AUC_{\tau, ss}$ | Area under the plasma concentration-time curve during a dose interval at steady state |
| b.i,d. | Twice daily |
| BLQ | Below limit of quantification |
| CDISC | Clinical data interchange consortium |
| CI | Confidence interval |
| $C_{\text{max, ss}}$ | Maximum plasma concentration at steady state |
| CSR | Clinical study report |
| $C_{trough, ss}$ | Trough plasma concentration at steady state |
| CV | Coefficient of variation |
| $CV_b$ | Inter-subject coefficient of variation |
| DBP | Diastolic blood pressure |
| ECG | Electrocardiograph |
| eCRF | Electronic case report form |
| EOS | End-of-study |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| IB | Investigator's Brochure |
| i.v. | Intravenous |
| ivSAF | intravenous Safety Analysis Set |
| LOQ | Limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MSE | Mean squared error |
| PAH | Pulmonary arterial hypertension |
| PDs | Protocol deviations |
| PK | Pharmacokinetic |
| PKS | Pharmacokinetic Analysis Set |
| PR | Pulse rate |

| Selexipag (ACT 293987) |
|-------------------------|
| Study AC-065A309 |
| 2 July 2018, page 7/135 |

# Confidential

Statistical Analysis Plan Doc No D-18.239

| PT | Preferred Term |
|---|---|
| QTcB | QT interval corrected using Bazett's formula |
| QTcF | QT interval corrected using Fridericia's formula |
| RMP | Risk Management Plan |
| SAE | Serious adverse event |
| SAF | Safety Analysis Set |
| SAP | Statistical analysis plan |
| $SAS^{\circledR}$ | Statistical Analysis Software |
| SBP | Systolic blood pressure |
| SCR | Screened Analysis Set |
| SD | Standard deviation |
| SDTM | Study data tabulation model |
| SE | Standard error of the mean |
| SOC | System organ class |
| $t_{\text{max, ss}}$ | Time to reach maximum plasma concentration at steady state |
| WHO | World Health Organization |
| WHO FC | WHO functional class |
| WHODD | WHO Drug Dictionary |

#### 1 INTRODUCTION

This statistical analysis plan (SAP) describes in detail the derivation of safety and pharmacokinetic (PK) endpoints and the analyses and the presentation of analysis results and data for the clinical study report (CSR) of study AC-065A309.

Study data tabulation model (SDTM) datasets, including data from central labs and PK data provided by Actelion Data Management will be considered source data. Technical procedures and steps for processing these data and for implementing the definitions of variables for the purpose of the statistical analysis in analysis data model (ADaM) datasets will be covered in the analysis datasets specifications document.

In this SAP, 'Uptravi®' refers to the prescribed presentation of oral selexipag; whereas 'i.v. selexipag' refers to the intravenous (i.v.) presentation of selexipag, which is considered the study drug.

This SAP is based on the following study documents:

Table 1 Study documents

| Document | Date, Version |
|---|---|
| Study Protocol | 27JAN2017, Version 1<br>19APR2017, Version 1.DEU.A (local) |
| eCRF specifications | 22SEP2017, Version 5 |
| Protocol deviation code list | 22FEB2017, Version 1.0 |
| Selexipag (Uptravi®) EU Risk Management Plan | 21JUN2017, Version 5.4 |
| ECG data transfer specification | 18AUG2017, Version 1.0 |
| Definition of Marked Abnormalities in Laboratory Data (OTH-000005) | 01NOV2017, Version 9 |

#### 2 STUDY DESIGN AND FLOW

# 2.1 Study design

This is a prospective, multi-center, open-label, single-sequence, cross-over, Phase 3 study.

Approximately 20 subjects with stable pulmonary arterial hypertension (PAH), currently treated with Uptravi (oral selexipag) at a stable dose, i.e., unchanged dose for at least 28 days, will be enrolled in order to obtain 18 evaluable subjects. Subjects will be stratified based on their stable Uptravi dose:

• Group A: Subjects with a stable dose of Uptravi between 200 and 1000 μg twice daily (b.i.d.) (inclusive); at least 5 and up to 8 subjects will be enrolled in this dose group.

• Group B: Subjects with a stable dose of Uptravi between 1200 and 1600 µg b.i.d. (inclusive); at least 12 and up to 15 subjects will be enrolled in this dose group.

The study will be conducted at approximately 10 sites in 2 countries.

# 2.2 Study visit and assessment schedule

The study visit and assessment schedule is included in Appendix A.

# 2.3 Analysis periods

The study comprises five analysis periods:

**Screening period:** This period starts with the signing of the Informed Consent Form and ends with the first day of Period 1 (Visit 2 Day 1).

**Period 1 (Uptravi, pre-treatment period, in-hospital):** This period starts with intake of the morning dose of Uptravi at Visit 2 Day 1, and ends the following day before initiation of the first infusion of i.v. selexipag.

**Period 2 (i.v. selexipag, treatment period, in-hospital):** This period starts in the morning of Visit 2 on Day 2 with the start of the first infusion of i.v. selexipag, and ends after approximately 36 hours in the evening of Visit 2 on Day 3 with the resuming of administration of Uptravi at the evening dose.

**Period 3 (Uptravi, post-treatment period):** This period starts in the evening of Visit 2 Day 3 with the first dose of resumed oral administration of Uptravi, and ends 7 to 11 days later at Visit 3.

**Safety follow-up period:** This period starts at the end of Visit 3 and ends 30 to 37 days after the last administration of i.v. selexipag with the End-of-Study (EOS) telephone call (Visit 4).

A summary of analysis periods is presented in Table 2:

Table 2 Summary of analysis periods

| Period | Start | Stop |
|---|---|---|
| Screening period | Date/time of first Informed consent form signature | Prior to morning dose of Uptravi at<br>Visit 2 Day 1 |
| Period 1:<br>Uptravi,<br>pre-treatment period | Date/Time of Uptravi morning dose intake at Visit 2 Day 1 | Prior to start of first infusion of i.v. selexipag at Visit 2 Day 2 |
| Period 2:<br>i.v. selexipag,<br>treatment period | Start date/time of first infusion of i.v. selexipag at Visit 2 Day 2 | Prior to evening dose of Uptravi at<br>Visit 2 Day 3 |
| Period 3:<br>Uptravi,<br>post-treatment period | Date/time of Uptravi evening dose intake at Visit 2 Day 3 | Visit 3 |
| Safety follow-up<br>period | After end of Visit 3 | End of Study |

The study design and flow is shown in Figure 1 below. For details, refer to section 3 and section 7 of the AC-065A309 study protocol [D-17.055].

Figure 1 Study design and flow



<sup>\* 12-</sup>hour PK profile after the morning dose.

<sup>\*\*</sup> For convenience, hospitalization may be extended to the night before Day 1 and to the night of Day 3.

D = day; EOS = End-of-Study; IV1-IV3 = dose of i.v. selexipag; PK = pharmacokinetic; V = visit.

# 2.4 Randomization and blinding

Not applicable, as this is a single-sequence, open-label study.

# 2.5 Sample Size

No confirmatory statistical tests are planned in the study.

Approximately 20 subjects will be enrolled to have at least 18 subjects in the i.v. Safety Set. In the GRIPHON Phase 3 pivotal study of selexipag, a proportion of 7.5% of subjects prematurely discontinued the study (i.e., without a morbidity/mortality event) due to prostacyclin-associated adverse events (AEs) across the titration and maintenance phases. It is expected that the proportion of early discontinuations during the entire study will not be higher than 10% (i.e., that approximately 18 subjects will enter the i.v. period).

A sample size of 18 subjects in the i.v. Safety Analysis Set will ensure that, if the true rate of discontinuations due to prostacyclin-associated AEs is between 5% and 10%, the half-width of the 95% confidence interval (CI) will be below 35%.

The precision achieved with a sample size of approximately 18 subjects in the i.v. Safety Set is considered adequate for this study (e.g., the upper boundary of the CI for the i.v. Safety Analysis Set excludes values above 35%, and for the Safety Analysis Set, above 32%).

#### 3 OBJECTIVES

# 3.1 Primary objective

The primary objective of this study is to assess whether temporary switching from a stable oral dose of selexipag to an i.v. dose of selexipag providing comparable exposure (e.g., area under the plasma concentration-time curve during a dose interval at steady state [AUC $_{\tau}$ , ss,], maximum plasma concentration at steady state [C<sub>max</sub>, ss]) to active metabolite ACT-333679 and switching back to the initial oral dose of selexipag is safe and well tolerated in subjects with stable PAH.

# 3.2 Other objectives

Other objectives of the study are:

- To evaluate the safety and tolerability of selexipag during each study period.
- To evaluate the PK of selexipag and its active metabolite, ACT-333679, at a stable oral dose at steady state and after the switch from selexipag oral to selexipag i.v. in subjects with stable PAH.

# 4 ANALYSIS SETS

# 4.1 Definitions of analysis sets

The following analysis sets were introduced in Section 10.1 of the protocol:

# 4.1.1 Screened Analysis Set

The **Screened Analysis Set** (SCR) includes all subjects who were screened and received a subject identification number.

# 4.1.2 Full Analysis Set

Not applicable in this study.

# 4.1.3 Safety Analysis Set

The Safety Analysis Set (SAF) includes all enrolled (included in the study on Day 1) subjects who received at least one dose of Uptravi or i.v. selexipag during any of Period 1, Period 2, or Period 3 of the study.

# 4.1.4 i.v. Safety Analysis Set

The i.v. Safety Analysis Set (ivSAF) includes all subjects who received at least one dose of i.v. selexipag.

# 4.1.5 Pharmacokinetic Analysis Set

The Pharmacokinetic Analysis Set (PKS) comprises all subjects included in the SAF who received an Uptravi dose on Day 1 and the three doses of i.v. selexipag, and who complied with the protocol in a way that the PK measurements of the study are not affected. Protocol deviations resulting in an exclusion from the PKS are shown in Table 3.

Additional rules for exclusion from the PKS may be defined prior to database lock and reflected in this document.

| Category | Protocol<br>deviation<br>code(s) | Identifier | Level of exclusion |
|---|---|---|---|
| Protocol deviation<br>during screening<br>period | 206 | Dose of Uptravi not stable for at least 28 days before Visit 2 (INCL 6) | Subject |
| | 209 | Subject with known and documented moderate and severe hepatic impairment (EXCL 2) | Subject |
| | 210 | Subject received gemfibrozil at any time since initiation of Uptravi (EXCL 3) | Subject |
| | 214 | Subject with renal failure and ongoing or planned dialysis (EXCL 7) | Subject |
| | 217 | Subject with another investigational treatment within 3 months of Visit 1 (EXCL 10) | Subject |
| Protocol deviation<br>during treatment and<br>observation period | 305 | Pre-dose PK blood sample collected after the morning dose on Day 1 or Day 3 | Data point* |
| | 306 | Any post-AM dose PK sample collected after administration of the following PM dose on Day 1 or Day 3 | Data point* |
| | 316 | Uptravi was not interrupted during i.v. selexipag treatment | Subject |
| | 312 | 25 min or 87 min post-infusion start PK blood sample on Day 3 collected from the same arm as the infusion line | Data point* |
| | 313 | Subject did not discontinue i.v. selexipag treatment despite missing one infusion | Subject |
| | 318 | Dose of PAH medications (including<br>diuretics) not stable between Visit 1<br>(screening) and last PK blood sample<br>collection on Day 3 | Subject |
| | 321 | Uptravi not administered or Uptravi dose missing on Day 1 | Subject |
| | 322 | Uptravi dose on Day 1 is different from stable dose at Visit 1 (screening) | Subject |
| | 323 | Any i.v selexipag dose is not corresponding to subject's stable dose of Uptravi (i.e., ≥ 225 ug)) | Subject |

<sup>\*</sup> If 2 or more data points are excluded from a 12-hour PK profile (i.e., on Day 1 or Day 3), the subjects must be excluded from the PKS. i.v. = intravenous; PK = pharmacokinetic; PKS = Pharmacokinetic Analysis Set.

# 4.2 Usage of the analysis sets

An overview on the usage of the analysis sets for summary tables and listings is given in Table 4.

Table 4 Overview of the different analysis sets and their usage

| Analyses/ Data Displays | Screened analysis set | Safety<br>analysis<br>set | i.v. Safety<br>analysis set | Pharmacokinetic analysis set |
|---|---|---|---|---|
| Demographic data (ICH E3 14.1) | | | | |
| Subject disposition | <b>✓</b> | <b>(</b> ✓)* | | |
| Protocol deviations | ✓ | | | |
| Inclusion/ Exclusion in Analysis<br>Sets | ✓ | | | |
| Subject characteristics<br>(Demographics, disease<br>characteristics, medical history) | | <b>✓</b> | | |
| Concomitant therapy | | ✓ | | |
| Study completion | | ✓ | | |
| Study treatment exposure and compliance | | ✓ | <b>√</b> ** | |
| PK data | | | | |
| PK endpoints, Period 1 & 2 | | | | ✓ |
| Safety data (ICH E3 14.3) | • | | | • |
| Adverse Events, Clinical Laboratory | y, ECG, Vital Sig | gns, Body Wei | ght and WHO FC* | :*<br>T |
| Period 1 | | ✓ | | |
| Period 2 | | | ✓ | |
| Period 3 | | | <b>√</b> | |
| Period 1 & 2 | | ✓ | | |
| Period 2 & 3& FU | | | ✓ | |
| Period 1 & 2 & 3 & FU | | ✓ | ✓ | |
| Appendices (ICH E3 16.1.7 and 16 All data collected in the clinical data | 6.2)<br>abase | | | |
| Listings | ✓ | ✓ | | |

<sup>\*</sup> Denominators for disposition will be based on the safety set. \*\* Tables will be produced for the SAF only if SAF and i.v. SAF are identical. ECG = electrocardiograph; FU = Safety Follow-Up; i.v. SAF = intravenous Safety Analysis Set; PK = pharmacokinetic; SAF = Safety Analysis Set; WHO FC = World Health Organization functional class.

#### 5 STUDY SUBJECTS VARIABLES AND ANALYSES

All summaries described in this section will be displayed separately for the two subject cohorts, i.e., subjects treated with Uptravi 200–1000  $\mu$ g b.i.d. and 1200–1600  $\mu$ g b.i.d., as well as for all subjects in the analysis set.

The summary tables, figures and listings will use the analysis sets shown in Table 4.

# 5.1 Subject disposition

The summaries of subject disposition and screening failures will be prepared on the SCR. Summaries of study completion/discontinuation and study treatment completion/discontinuation will be prepared on the SAF:

# 5.1.1 Subject disposition and enrollment into analysis periods

Subject disposition will be summarized by presenting the number of subjects screened, enrolled and then number and percentage of subjects entering each analysis period [see Section 2.3], number and percentage of subjects treated with one, two, and three doses of i.v. selexipag as well as the number and percentage of subjects completing or discontinuing i.v. treatment or the study.

In addition, a summary of disposition by site and country will be prepared.

# 5.1.2 Screening failures

Screening failures are subjects who were not enrolled into the study, i.e., subjects who did not enter Period 1 of the study.

The number of screening failures will be shown in the disposition table. Reasons for screening failure will be listed.

#### 5.1.3 Study completion/discontinuation

Subjects who received at least one dose of i.v. selexipag and who have completed the follow-up period will be considered study completers.

Subjects may discontinue from the study by withdrawal of consent, loss to follow-up, death, or investigator or sponsor decision. Details of study discontinuation are collected in the electronic case report form (eCRF).

The number and percentages of subjects who completed or prematurely discontinued the study, and reasons for discontinuation from the study will be summarized in a table and in a listing.

# 5.1.4 Study treatment completion/discontinuation

The number and percentage of subjects who completed or prematurely discontinued i.v. selexipag treatment, and reasons for premature discontinuation from i.v. selexipag treatment as captured in the eCRF will be summarized in a table and in a listing.

#### 5.2 Protocol deviations

The analysis of protocol deviations (PDs) will be prepared on the SCR.

PDs will be based on the PD code list. The PD code list may be updated during the course of the study, but before database closure. The number and percentage of subjects who had an important PD will be summarized overall. All PDs will be summarized overall and by country.

All PDs will be listed. This listing includes all deviation descriptions, identifiers and categories.

# 5.3 Exclusion from analysis sets

The number and percentage of subjects in each analysis set, as described in Section 4.1, will be summarized in a table together with the number and percentage of subjects excluded from any analysis set, together with the reasons for exclusion. A listing of subject participation in the different analysis sets will be produced.

# 5.4 Subject characteristics

Subject characteristics will be summarized on the SAF.

#### 5.4.1 Demographics

Baseline demographics, body weight and height will be summarized. The summary will include:

- Age (years)
- Sex (categorized as: Male, Female)
- Race (categorized as: American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or other Pacific Islander, White, Other)
- Ethnicity (categorized as: Hispanic or Latino, Not Hispanic or Latino, Unknown)
- Body weight (kg)
- Height (cm)
- Country (assigned in the eCRF based on the list of sites).

In addition, the following variables will be derived:

- Age (years) in category, i.e., > = 18 < 65, > = 65 years
- Body mass index (kg/m<sup>2</sup>)

Demographic characteristics will be summarized using descriptive statistics for continuous and categorical data. Demographic characteristics will also be listed.

For disclosure of results to EudraCT, a summary table will be created showing age (years) in categories 18-64, 65-84, and > = 85.

#### **5.4.2** Baseline disease characteristics

Baseline disease characteristics comprise the specific medical history (time since the initial diagnosis of PAH, and etiology of PAH as well as Uptravi dose) assessed at the screening visit and the WHO functional class (WHO FC) at Day 1.

Baseline disease characteristics will be summarized using descriptive statistics for continuous and categorical data. Time since initial diagnosis of PAH will be summarized in months.

Baseline disease characteristics will be listed.

#### **5.4.3** Other baseline characteristics

The results of a physical examination will be listed.

#### 5.4.4 Medical history

Medical history includes relevant previous and/or concomitant diseases or diagnoses prior to or ongoing at Screening visit, respectively. They are recorded on the 'Medical History' eCRF page. Reported terms will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at database lock, Version 21.0.

**Previous diseases or diagnoses** are medical history events which are not ongoing at screening, i.e., they have an end date prior to or equal to the Screening visit.

Concomitant diseases or diagnoses are all medical history events that are not considered as previous events.

Previous and concomitant diseases/diagnoses will be summarized separately by tabulating the number and percentages of subjects with each disease/diagnosis by system organ class (SOC) and preferred term (PT).

Previous and concomitant medical diseases/diagnoses will be listed.

#### 5.4.5 Previous and concomitant therapies

Previous and concomitant therapies are collected continuously in the eCRF. The reported names will be coded using the WHO drug code dictionary (WHODD) and the anatomic therapeutic chemical (ATC) class code.

**Previous therapies** are therapies which ended prior to baseline [see Section 10.2].

**Ongoing therapies** are therapies that were started prior to baseline and are ongoing at study treatment start.

**Study concomitant therapies** are therapies that were started or dose changed (of those ongoing at baseline) during the respective analysis period [see Table 2].

Previous therapies, ongoing therapies, and study concomitant therapies will be summarized separately by Level 4 ATC class and PT. The study concomitant therapies summary will be displayed by study period.

The summaries will exclude PAH-specific therapies [see Section 5.4.5.1].

All recorded terms will be reported together in one listing together with flags indicating the type of therapy.

# 5.4.5.1 PAH-specific therapies

PAH-specific therapies will be identified by a search of WOHDD PTs and ingredients as shown in Table 5. Specific summaries will be prepared:

Ongoing PAH-specific therapies at baseline will be summarized. PAH-specific therapies that are newly started, dose changed, or stopped during any study period will be listed in a separate listing.

PAH-specific therapies will be displayed in a listing with the respective study period flagged.

Table 5 PAH-specific therapies

| Category | Subcategory | Ingredient names |
|---|---|---|
| Antihypertensives for pulmonary arterial hypertension | ERAs | Ambrisentan, Bosentan, Macitentan |
| | PDE-5 inhibitors | Sildenafil, Tadalafil, Vardenafil |
| | sGC stimulator | Riociguat |
| Prostanoids | | Epoprostenol, Treprostinil, Iloprost, |
| Uptravi | | Selexipag |

Categories are identified by searching the coded WHODRUG preferred terms for occurrence of any of the ingredient names, e.g., 'Sildenafil' and 'Sildenafil Citrate' will both be assigned to PDE-5 inhibitors.

ERA = endothelin receptor antagonist; PAH = pulmonary arterial hypertension; PDE-5 = phosphodiesterase type-5; sGC = soluble guanylate cyclase.

#### 5.4.5.2 Auxiliary medications

Oral Uptravi is collected as a mandatory background drug in the previous and concomitant medication page. Dose changes will be listed with PAH-specific therapies.

# 5.5 Study treatment exposure and compliance

i.v. selexipag is considered the only study treatment for this study.

#### 5.5.1 Exposure

#### 5.5.1.1 Exposure to i.v. selexipag

The number and percentage of subjects being exposed to one, two, or three infusions of i.v. selexipag will be summarized.

The planned i.v. selexipag dose  $[\mu g]$  for each infusion will be summarized as a continuous variable as well as a categorical variable using categories from Table 6. The actual i.v. selexipag dose will be summarized separately. Total actual time of infusion in minutes will be summarized for each of the three infusions as well.

The summary will be conducted for each of the three infusions separately.

The dosage administration records will be listed together with the reasons for dose change and dosage end as recorded in the eCRF.

# 5.5.1.2 Exposure to Uptravi prior and post- i.v. selexipag

The actual Uptravi dose  $[\mu g]$  will be collected and summarized by dose category for the four time points surrounding the i.v. administration of selexipag, i.e., evening dose before Visit 2 Day 1, morning and evening dose at Visit 2 Day 1 and evening dose at Visit 2 Day 3.

The Uptravi dosage records will be listed.

# 5.5.1.3 Shift in selexipag dose between oral and i.v. treatment

The shift from actual oral to i.v. and back to oral doses will be analyzed graphically in a series plot showing the individual dose in  $[\mu g]$  for each dose administration time point during Day 1 through Day 3 of Visit 2.

The i.v. selexipag doses administered will be converted to their oral dose equivalents [see Table 6] to facilitate the review.

# 5.5.1.4 Study treatment adjustments or interruptions, end of infusion status

Incidence of and reasons for i.v. administration interruption as well as the end of infusion status (irrespective of whether study treatment was completed as per protocol or not) will be summarized for each of three infusions.

# 5.5.2 Compliance with study treatment

Compliance with i.v. selexipag treatment is defined as the percentage of the actual dose infused compared with the planned dose to be infused, for each infusion and overall.

The planned dose to be infused will be determined from Table 6 below and based on the subjects' stable Uptravi dose taken from the Visit 2 Day 1 evening dose.

Table 6 Correspondence of i.v. selexipag dose compared to Uptravi oral doses

| Uptravi oral dose (µg) | Corresponding i.v. selexipag dose (μg) |
|------------------------|----------------------------------------|
| 200 | 225 |
| 400 | 450 |
| 600 | 675 |
| 800 | 900 |
| 1000 | 1125 |
| 1200 | 1350 |
| 1400 | 1575 |
| 1600 | 1800 |

The actual infused dose will be computed by computing the product of the infusion rate (mL/h) with the concentration of infusion solution  $(\mu g/mL)$  as recorded in the eCRF and the elapsed time between start and end time (h) for each infusion to obtain the amount of i.v. selexipag infused.

Missed infusions will be entered with 0 µg actual infusion into the compliance analysis.

The planned dose, actual dose, and resulting compliance will be listed. Compliance will be summarized descriptively for each period and overall.

#### 6 EFFICACY VARIABLES AND ANALYSES

Not applicable in this study.

#### 7 SAFETY VARIABLES

#### 7.1 Overview of safety analyses including subgroup analyses

# 7.1.1 Overview of safety and tolerability endpoints

Safety endpoints in this study comprise the incidence of AEs and serious AEs (SAEs), discontinuations due to AEs, change and newly occurring abnormalities in vital signs, ECG and clinical laboratory values, as well as change in WHO FC and body weight.

The analysis of safety endpoints in different analysis periods [see Table 2] is summarized in Table 7 below.

Table 7 Overview of safety and tolerability endpoints and populations in planned analysis periods

| Endpoint | SCR<br>(Scr) | 1<br>(S) | 2<br>(ivS) | 3&FU<br>(ivS) | 1&2<br>(S) | 2&3&FU<br>(ivS) | 1&2&3&FU<br>(S, ivS) |
|---|---|---|---|---|---|---|---|
| Main safety and tolerability endpoints | | | | | | | |
| AEs and SAEs | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Prostacyclin-associated AEs <sup>1</sup><br>leading to discontinuation of study<br>drug | | | ✓ | | | | |
| Prostacyclin-associated AEs1 | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Injection site reaction AEs <sup>1</sup> | | | ✓ | | | | |
| PAH related AEs <sup>1</sup> | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Other safety and tolerability endpoints | | | | | | | |
| AEs leading to discontinuation of study drug | | | ✓ | | | | |
| AEs related to study drug as judged by the investigator | | | ✓ | ✓ | | ✓ | ✓ |
| Deaths during study | | | | | | | ✓ |
| ECG abnormalities, QT prolongation | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Marked laboratory abnormalities | | ✓ | ✓ | ✓ | | ✓ | ✓ |
| Marked blood pressure abnormalities | | ✓ | ✓ | ✓ | | ✓ | ✓ |
| Change from baseline in WHO functional class <sup>2</sup> | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |

Periods connected by an ampersand will be analyzed combined.

All analyses will be run on the S, if S and ivS are identical.

<sup>&</sup>lt;sup>1</sup> As defined by MedDRA search terms <sup>2</sup> By visit analyses

<sup>(</sup>S) = Safety analysis Set, (ivS) = i.v. Safety analysis set, (Scr) = Screened subject set; AE = adverse event; ECG = electrocardiograph; FU = Safety Follow Up; MedDRA = Medical Dictionary for Regulatory Activities; PAH = pulmonary arterial hypertension; SAE = serious adverse event; SCR = Screening period, WHO = World Health Organization.

#### 7.2 Adverse events

#### 7.2.1 Variables

The original verbatim terms used by investigators to identify AEs in the eCRF will be mapped to PTs using the MedDRA dictionary using the latest version at data cutoff. The AE PTs will be then grouped by MedDRA PTs into frequency tables according to primary SOC.

# 7.2.1.1 Treatment-emergent adverse events

The analysis of AEs in Period 2, Period 3 and safety follow-up period is considered analysis of treatment-emergent events, as the i.v. formulation is the investigational treatment.

# 7.2.1.2 Adverse events related to study treatment

An AE will be considered related to the study treatment if the investigator answered 'yes' to the question 'Causal relationship to i.v. selexipag' or if it is missing.

# 7.2.1.3 Serious adverse events

An AE will be considered serious if the investigator answered 'Yes' to the question 'Serious?' or if information is missing.

# 7.2.1.4 Adverse events leading to discontinuation of study treatment

An AE is considered as leading to discontinuation of study treatment if the investigator ticked 'Drug withdrawn' on the question 'Action taken with study treatment'.

#### 7.2.1.5 Injection site reactions

Injection site reactions will be collected on a separate eCRF page. Clinically significant injection site reactions will be reported as an AE.

#### 7.2.1.6 Prostacyclin-associated AEs

Prostacyclin-associated AEs are AEs associated with the pharmacological action of selexipag that have been observed frequently, in particular during the phase of individualized dose titration. According to selexipag Investigator's Brochure (IB) reference safety information, these PTs include headache, diarrhea, nausea, vomiting, jaw pain, myalgia, pain in the extremity, flushing, and arthralgia.

# 7.2.1.7 AEs of special interest based on the Uptravi Risk Management Plan

For completeness, AEs will be analyzed according to the Uptravi Risk Management Plan (RMP) important identified or potential risks, using searches of MedDRA PTs provided by Global Drug Safety at the time of database closure. In accordance with the RMP, the following categories will be analyzed:

- Hypotension
- Anemia, decrease in hemoglobin concentration

Statistical Analysis Plan Doc No D-18.239

- Hyperthyroidism
- Major adverse cardiovascular events
- Acute renal failure
- Bleeding events
- Light-dependent non-melanoma skin tumors
- Ophthalmological effects associated to retinal vascular system
- Gastrointestinal disturbances denoting intestinal intussusception (manifested as ileus or obstruction).

# 7.2.1.8 PAH-related AEs

PAH-related AEs are AEs that are coded to the following MedDRA (Version 21.0) PTs:

Atrial fibrillation Lung transplant

Atrial flutter Pulmonary arterial hypertension

Atrial natriuretic peptide abnormal Pulmonary arterial pressure abnormal

Atrial natriuretic peptide increased Pulmonary arterial pressure increased

Acute right ventricular failure Pulmonary oedema

Cardiac failure Pulmonary hypertension

Cardiac index decreased Pulmonary hypertensive crisis

Cardiogenic shock Right atrial dilatation

Cardiopulmonary failure Right atrial pressure increased

Chronic right ventricular failure Right ventricular dysfunction

Cor pulmonale Right ventricular failure

Cor pulmonale acute Syncope

Oedema peripheral Vascular resistance pulmonary increased

Jugular vein distension

#### 7.2.1.9 Non-serious AEs

For the disclosure of the results to EudraCT and ClinicalTrials.gov, non-serious AEs are defined. A non-serious AE is any AE with the question "Serious?" answered "No" by the investigator.

#### 7.2.2 Analysis

The start date/time of the AE record from the CRF will be used to assign the AE to a study period.

Summary tables will be prepared as described in Table 8 for the periods mentioned in Table 7, except for the screening period.

Summary tables by SOC and PT will display the number and percentages of subjects with at least one AE in the respective primary SOC and at least one AE at the PT level. Summaries will be sorted by descending total frequency of SOCs and PTs and alphabetically in case of ties.

Summary tables by PT will display the number and percentages of subjects with at least one AE in the respective PT. Summaries will be sorted by descending total frequency of PTs and alphabetically in case of ties.

AEs occurring during the Screening period, i.e., prior to first dose of Uptravi on Visit 2 Day 1, will be listed.

Due to the small number of subjects, conservative 95% Clopper-Pearson CIs for the proportions will be computed using exact methods.

All AEs occurring during the study from date of informed consent signature to EOS will be listed.

For any injection site reaction (irrespective of clinical significance), the worst grade, criteria of the injection site reaction, as well as its clinical significance will be summarized. Any AEs associated with clinically significant injection site reactions will be summarized by PT and by maximum intensity in the AE table.

| Category | Approach |
|---|---|
| All AEs | <ul> <li>N (%) of subjects having at least one AE by primary SOC and PT</li> <li>N (%) of subjects having at least one AE by PT</li> <li>N (%) of subjects having at least one AE by PT and maximum intensity</li> <li>Listing</li> </ul> |
| SAEs | - N (%) of subjects having at least one SAE by PT - Listing |
| Injection site reaction AEs | <ul> <li>N(%), grade and diagnosis criteria of injection site reactions</li> <li>N (%) of subjects having at least one clinically significant injection site reaction by PT and maximum intensity</li> <li>Listing of PTs and specific details</li> </ul> |
| Prostacyclin-associated AEs | <ul> <li>N (%) of subjects having at least one prostacyclin associated AE by PT</li> <li>N % of subjects having at least one prostacyclin associated SAE by PT</li> <li>N % of subjects having least one prostacyclin associated AE leading to discontinuation of study drug by PT</li> <li>Listing</li> </ul> |
| AEs of special interest based on<br>the Uptravi RMP | <ul> <li>N (%) of subjects having at least one AE by RMP category and PT</li> <li>N % subjects having at least one SAE by RMP category and PT (Listing)</li> <li>N % least one AE by RMP category leading to discontinuation of study drug by RMP category and PT</li> <li>Listing</li> </ul> |
| PAH-related AEs | - N (%) of subjects having at least one event by PT - Listing of events |
| Any AE leading to discontinuation of study drug | - N (%) of subjects having at least one event by PT - Listing of events |
| AEs related to study drug as judged by the investigator | - N (%) of subjects having at least one event by PT - Listing of events |

AE = adverse event; PAH = pulmonary arterial hypertension; PT = Preferred Term; RMP = Risk Management Plan; SAE = serious adverse event; SOC = System Organ Class.

# 7.2.2.1 Summaries of adverse events for public disclosure

For the disclosure of the results to EudraCT and ClinicalTrials.gov (and not for the purpose of the clinical study report), treatment-emergent (S)AEs will be summarized displaying, for each dose group, counts and percentages of subjects with at least one treatment-emergent event plus the number of events (counted exactly the number of times they occurred also within a subject) by SOC and individual PT. The summary table is presented in descending order according to the overall incidence (i.e., SOC and

individual PT within each SOC with the highest number of occurrences appears first). Equal frequency of different individual PTs is sorted in alphabetical order of the individual PT.

The following summaries will be prepared according to the guidelines stated above:

- Summary of treatment-emergent SAEs
- Summary of treatment-emergent SAEs judged to be treatment related by the investigator
- Summary of treatment-emergent SAEs with fatal outcome
- Summary of treatment-emergent SAEs with fatal outcome judged to be treatment related by the investigator
- Summary of non-serious AEs with an incidence of 5% or higher in any treatment group

#### 7.3 Deaths

Date of death and primary cause will be recorded on the 'Death' eCRF page. A listing including all deaths recorded in the database will be provided.

A separate listing will be provided displaying all AEs leading to death, i.e., with outcome 'fatal'.

# 7.4 Laboratory

A central laboratory will be used for all protocol-mandated tests. Laboratory values analyzed by local laboratories will only be listed.

Laboratory test results will be converted into Standard International units by the laboratory. Values outside the laboratory normal ranges will be flagged as well.

#### 7.4.1 Measurements

Laboratory test results will be transferred from the central laboratory and provided in the SDTM structure, together with corresponding reference ranges in original, conventional, and standardized units. Assessments are performed at Screening visit, Visit 2 Day 1 (if more than 7 days after screening), Visit 2 Day 3, Visit 3, and at unscheduled visits based on the judgment of the investigator.

The following variables are collected as per protocol:

#### Hematology

- Hemoglobin (g/L)
- Hematocrit (L/L)
- Erythrocytes (10<sup>12</sup>/L)

- Leukocytes with differential counts (10<sup>9</sup>/L)
- Platelets (10<sup>9</sup>/L)

# **Clinical chemistry**

- Alanine aminotransferase (ALT) (U/L)
- Aspartate aminotransferase (AST) (U/L)
- Alkaline phosphatase (AP) (U/L)
- Total and direct bilirubin (μmol/L)
- Creatinine (µmol/L)
- Sodium, potassium (mmol/L)

For women of childbearing potential, urine pregnancy tests are performed at Screening Visit, Visit 2 Day 1, and Visit 4 (EOS). A pregnancy will be reported as an SAE; the results of the pregnancy tests will not be included in the clinical database.

#### 7.4.2 Variables

For parameters assessed as a continuous variable, the following variables will be defined:

- Baseline
- Value at each post-baseline visit
- Absolute change from baseline to each post-baseline visit
- Position against reference ranges based on normal ranges provided by the laboratory.
- Position against marked abnormality range based on ranges provided in Appendix D.

#### 7.4.3 Analysis

All laboratory values will be listed. Values from local laboratories will be flagged in data listings and not used in any analysis.

#### 7.4.3.1 Values over time

For continuous laboratory variables, descriptive statistics will be provided for observed values as well as for change from baseline at each scheduled study visit.

#### 7.4.3.2 Individual subject changes

Laboratory test results from both, scheduled and unscheduled visits will be used to determine the incidence of markedly abnormal test results. The date of the sample will determine the analysis period the test is assigned to.

The number of subjects with newly occurring or worsening markedly abnormal laboratory values will be displayed for the analysis sets shown in Table 4 and the periods shown in Table 7.

The definitions of marked abnormal lab values are shown in Appendix D.

# 7.5 Vital signs, physical findings, and other observations related to safety

# 7.5.1 Vital signs

Vital signs will be collected in an eCRF. Systolic blood pressure (SBP) and diastolic blood pressure (DBP) and pulse rate (PR) assessed in supine position will be entered in mmHg. Height (cm) and weight (kg) will be assessed in subject wearing indoor clothing without shoes.

#### 7.5.1.1 Measurements

Height (cm) will be assessed at Screening Visit.

Body weight will be assessed at Screening visit, Visit 2 Day 1, Visit 2 Day 3, Visit 3 and at unscheduled visits.

SBP, DBP, and PR will be assessed at Screening visit, Visit 2 Day 1, Visit 3 and at unscheduled visits. Further assessments will be conducted at pre-specified time points in Period 2, i.e., Visit 2 Day 1 and Visit 2 Day 3 as shown in Table 9.

Table 9 Schedule vital signs monitoring in Period 2

| Visit Day | Time point | Assessment Description |
|---|---|---|
| Visit 2 Day 2 | 0 h | Shortly before morning (AM) i.v. selexipag infusion |
| | 25 min | During AM i.v. selexipag infusion, 25 min after infusion start |
| | 87 min | Shortly before end of AM i.v. selexipag infusion |
| | 4 h | Four hours after initiation of AM selexipag infusion |
| | 6 h | Six hours after initiation of AM selexipag infusion |
| | 8 h | Eight hours after initiation of AM selexipag infusion |
| | 12 h | Before PM selexipag infusion,<br>twelve hours after initiation of AM selexipag infusion |
| Visit 2 Day 3 | 0 h | Shortly before morning (AM) selexipag infusion |
| | 25 min | During AM selexipag infusion, 25 min after infusion start |
| | 87 min | Shortly before end of AM selexipag infusion |
| | 4 h | Four hours after initiation of AM selexipag infusion |
| | 6 h | Six hours after initiation of AM selexipag infusion |
| | 8 h | Eight hours after initiation of AM selexipag infusion before oral administration of selexipag |
| | 12 h | Before PM Uptravi intake,<br>twelve hours after initiation of AM selexipag infusion |

# 7.5.1.2 Variables

For vital signs parameters, the following variables will be defined:

- Baseline
- Value at each post-baseline visit
- · Absolute change from baseline to each post-baseline visit
- Absolute change from pre-dose to each post-dose assessment.

For supine SBP (mmHg) and supine DBP (mmHg), the presence of post-baseline abnormalities is derived according to the criteria defined in Table 10 below:

Table 10 Marked abnormalities in blood pressure

| Analysis<br>Parameter | LL | L | Normal | H | нн |
|---|---|---|---|---|---|
| Supine SBP (mmHg) | - | SBP < 90 | 90 ≤ SBP < 140 | $140 \le SBP \le 159$ | $SBP \geq 160$ |
| | - | Decrease > 40 from baseline | - | Increase > 20 from baseline | - |
| Supine DBP (mmHg) | - | DBP < 50 | 50 ≤ DBP < 90 | $90 \le DBP \le 99$ | $DBP \geq 100$ |
| | - | Decrease > 20 from baseline | - | Increase > 20 from baseline | - |

DBP = diastolic blood pressure; SBP = systolic blood pressure.

Abnormalities will be flagged for each post-baseline assessment individually and overall for the study treatment period.

# 7.5.1.3 *Analysis*

#### Values over time

A listing of all vital sign parameters will be created displaying all values in the database regardless if from scheduled or unscheduled visits. Marked abnormal values will be flagged.

Descriptive statistics will be provided for observed values as well as for change from baseline to all visits.

Another descriptive summary will be provided for the absolute change from pre-dose to post-dose values for the visits where pre- and post-dose values are assessed.

#### Individual subject changes

The number and percentage of subjects with at least one marked newly occurring or worsening abnormality for blood pressure will be summarized by period (Period 2, Period 3/ Safety follow-up [FU]) and overall (Period 2, 3, and FU combined) as shown in Table 7.

# 7.5.2 Physical findings

Physical examination will be conducted at screening, may be repeated at Visit 2 Day 1, and will be conducted at Visit 3.

The results of the physical examination will be listed. New abnormal physical findings will be reported as AEs.

#### 7.5.3 WHO functional class

WHO FC (Class I–IV) as assessed by the investigator will be collected in the eCRF.

#### 7.5.3.1 Measurements

WHO FC will be assessed at Screening Visit, Visit 2 Day 1, Visit 2 Day 3 (after the end of the last infusion), Visit 3, and at unscheduled visits.

#### 7.5.3.2 Variables

For WHO FC, the following variables will be defined:

- Baseline value
- Value at each post-baseline visit
- Shift from baseline to each post-baseline visit
- Worst (highest) post-baseline value
- Best (lowest) post-baseline value.

# 7.5.3.3 *Analysis*

#### Values over time

A listing of all WHO FC assessments will be created displaying all values in the database, regardless if from scheduled or unscheduled visits.

Descriptive statistics (frequency tables) will be provided for observed values as well as for shift from baseline to all visits.

#### Individual subject changes

The worst/best post-baseline WHO FC will be displayed along with a shift table from baseline to worst/best post-baseline value.

# 7.6 Electrocardiograph

A standard 12-lead electrocardiograph (ECG) will be conducted on subjects in fully rested supine position. All ECG data from scheduled and unscheduled visits will be transferred to a central ECG laboratory. The ECG readouts (see below) will be transferred from the central ECG laboratory to trial data management and imported in the trial database.

#### 7.6.1 Variables

The 12-lead ECG encompasses 3 categories of data obtained via the central ECG laboratory:

- Measurements:
  - ECG mean heart rate
  - PR interval,
  - QRS duration,
  - QT interval,
  - QTcB interval,
  - QTcF interval,
- Interpretation (normal/abnormal/unable to evaluate)
- Qualitative findings by category, as specified in the ECG data transfer specifications:

# Table 11 Pre-specified ECG findings categories

| Category |
|-----------------------------------------|
| Atrioventricular Conduction |
| Axis and Voltage |
| Chamber Hypertrophy or Enlargement |
| Intraventricular-Intraatrial Conduction |
| Myocardial Infarction |
| Pacemaker |
| Sinus Node Rhythms and Arrhythmias |
| Supraventricular Arrhythmias |
| Supraventricular Tachyarrhythmias |
| ST Segment, T Wave and U wave |
| Ventricular Arrhythmias |
| Ventricular Tachyarrhythmias |

ECG assessments will be performed at Visit 2 Day 1, Visit 2 Day 2 (pre-dose and 30 min after end of infusion for each of the two infusions), Visit 2 Day 3 (pre-dose and 30 min after end of infusion), Visit 3, and at unscheduled visits.

#### 7.6.2 Variables

The following variables will be defined for the analysis of ECG parameters:

- Baseline values of quantitative ECG parameters
- Value at each post-baseline visit
- Absolute change from baseline to each post-baseline visit
- Absolute change from pre-dose after each infusion
- Proportion of qualitative ECG abnormalities

In addition, the incidence of QT prolongations is derived according to the criteria defined in Table 12 below:

Table 12 QT prolongations in ECG parameters

| Analysis Parameter | Analysis Variable(s) | Analysis Criterion |
|---|---|---|
| QTcB (msec)<br>QTcF (msec) | Analysis value | - Value > 450<br>- Value > 480<br>- Value > 500 |
| | Change from baseline | <ul><li>Increase from baseline &gt; 30</li><li>Increase from baseline &gt; 60</li></ul> |
| | Analysis value and change from baseline | <ul> <li>Value &gt; 450 and increase from baseline &gt; 30</li> <li>Value &gt; 450 and increase from baseline &gt; 60</li> </ul> |

ECG = electrocardiograph; QTcB = QT interval corrected using Bazett's formula;

QTcF = QT interval corrected using Fridericia's formula.

# 7.6.3 Analysis

#### 7.6.3.1 Values over time

A listing of all ECG measurements will be created displaying all values in the database. Abnormal ECG values will be flagged.

The overall interpretation and the findings will be presented in a separate listing.

For each parameter at each time over the course of the study, quantitative descriptive statistics for the value at the visit and the change from baseline will be presented by parameter and by time point.

Another descriptive summary will be provided for the absolute change from pre-dose to post-dose values in quantitative ECG parameters for the visits where pre- and post-dose values are assessed.

#### 7.6.3.2 Individual subject changes

The number and percentage of subjects with at least one newly occurring or worsening abnormality for ECG parameters as defined in Table 12 is provided by period as shown in Table 7.

In addition, qualitative ECG findings will be tabulated by overall interpretation (normal, abnormal/unable to evaluate), and category [see Table 11].

# 7.7 Subgroup analysis of safety variables

In general, all safety variable summaries are presented by dose cohort as for study subject analyses [see Section 5].

No *a-priori* subgroup analyses are planned at this point.

#### 7.8 Pharmacokinetic variables

#### 7.8.1 Measurements

PK blood samples are collected at Visit 2 Day 1 (seven samples) and Visit 2 Day 3 (seven samples) to obtain 12-hour PK profiles of selexipag and its active metabolite, ACT-333679, at steady state for Uptravi and i.v. selexipag, respectively.

Endpoints derived during Period 1 are thus connected to Uptravi (Day 1) and endpoints during Period 2 are connected to i.v. selexipag (Day 3).

# 7.8.2 Pharmacokinetic endpoints

The following PK endpoints will be determined:

- AUC<sub> $\tau$ , ss</sub> of selexipag and its active metabolite, ACT-333679, after Uptravi (oral selexipag) in Period 1 and after i.v. selexipag administration in Period 2.
- C<sub>max, ss</sub> of selexipag and its active metabolite, ACT-333679, after Uptravi (oral selexipag) in Period 1 and i.v. selexipag administration in Period 2.
- The time to reach maximum plasma concentration at steady state (t<sub>max, ss</sub>) of selexipag and its active metabolite, ACT-333679, after Uptravi (oral selexipag) in Period 1 and i.v. selexipag administration in Period 2.
- Trough plasma concentration at steady state (C<sub>trough, ss</sub>) of selexipag and its active metabolite, ACT-333679, after Uptravi (oral selexipag) in Period 1 and i.v. selexipag administration in Period 2.

#### 7.8.3 Pharmacokinetic variables

Plasma PK parameters of selexipag and its active metabolite, ACT-333679, will be derived by non-compartmental analysis of the concentration-time profiles.

The PK parameters will be calculated on the basis of the real blood sampling time points (in relation to the last selexipag intake during each period).

The measured individual plasma concentrations of selexipag will be used to directly obtain  $C_{trough, ss}$ ,  $C_{max, ss}$ , and  $t_{max, ss}$ .

 $AUC_{\tau, ss}$  will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ) during one dosing interval at steady state.

# 7.8.3.1 Dose normalization

Dose normalization will be conducted to the lowest prescribed selexipag dose (200 µg for oral Uptravi and 225 µg for i.v. selexipag).

Dose normalized plasma concentrations,  $C_{trough, ss, norm}$ ,  $C_{max, ss, norm}$  and  $AUC_{\tau, ss, norm}$  will be determined by dividing the respective parameters by the actual dose and multiplying with 200 or 225 for Uptravi and i.v. selexipag parameters, respectively.

# 7.8.4 Analysis

All PK parameters will be listed for all subjects providing PK data. All analyses will be conducted on the PKS.

For mean value calculations, all values below the limit of quantification (BLQ) will be set to zero. If > 50% of the values at a given time point are BLQ, no mean value will be calculated. Mean concentration-time profiles will be generated using these criteria.

#### 7.8.4.1 Plasma concentrations

The PK expert will examine the plasma concentration data and identify implausible values.

Plasma concentrations of selexipag and ACT-333679 will be listed per subject, time point, and period (i.e., for Uptravi and i.v. selexipag). Implausible plasma concentrations of selexipag or ACT-333679 will be flagged in the listings.

Plasma concentrations of selexipag and ACT-333679 will be summarized per time point by dose, including dose normalized, and period (i.e., for Uptravi and i.v. selexipag). Implausible plasma concentrations of selexipag or ACT-333679 will not be included in the summary statistics.

Implausible values will be indicated in the comments value variable (COVAL) of the comments dataset (CO). The reference link (COREF) will be used to join these implausible values with time points of the plasma concentration dataset (PC).

#### 7.8.4.2 Trough concentrations

Selexipag and ACT-333679 C<sub>trough, ss</sub> will be listed by dose, subject, and period as well as the ratio of the periods per subject.

Summary statistics will be provided by dose, including dose normalized, and by period. Implausible  $C_{trough, ss}$  values will be flagged in the listings and not included in summary statistics.

# 7.8.4.3 $C_{max, ss}$ , $t_{max, ss}$ , and $AUC_{\tau, ss}$

 $C_{max, ss}$ ,  $t_{max, ss}$ , and  $AUC_{\tau, ss}$  of selexipag and ACT-333679 will be listed by dose, subject, and period. The ratio of the parameters between i.v. selexipag (test treatment) and Uptravi (reference treatment) per subject will be shown, except for  $t_{max, ss}$ . Any values

obtained from implausible plasma concentrations of selexipag or ACT-333679 will be flagged in the listings and not included in the statistical analysis.

Summary statistics will be provided by dose and period for selexipag and ACT-333679.

Dose-normalized  $C_{max, ss}$  and  $AUC_{\tau, ss}$  will be listed and summarized by period as well for selexipag and ACT-333679.

 $C_{max, ss}$  and  $AUC_{\tau, ss}$  ratio of ACT-333679/selexipag will be listed by dose, subject, and treatment and will be summarized by dose and treatment.

The ratio of  $C_{max, \, ss}$  and  $AUC_{\tau, \, ss}$  of selexipag and ACT-333679 between Uptravi and i.v. selexipag, after dose normalization, within each dose level (if sufficient subjects are enrolled per level) will be estimated by fitting a mixed effect model to the data using period (i.e., treatment) as fixed, and subject as random effect to the log-transformed  $C_{max, \, ss}$  and  $AUC_{\tau, \, ss}$  values. The ratios of geometric means between i.v. selexipag (test treatment) and Uptravi (reference treatment) will be computed and displayed together with their 90% CI by back-transforming the period contrasts and interval boundaries of the log-transformed data. If dose-proportionality is shown within each dose, then an overall model may be considered for robustness.

The inter-subject coefficient of variation (CV<sub>b</sub>) of  $C_{max, ss}$  and  $AUC_{\tau, ss}$  of selexipag and ACT-333679 will be computed by using the mean squared error (MSE) of the mixed model as an estimate of variation.

Based on the previous studies QGUY/2006/NS304/-01, AC-065-101 and AC-065A201 it is known that the PK profile of selexipag and its active metabolite ACT-333679 is dose-proportional up to a single dose of 800 ug and for multiple doses of up to 1800 ug b.i.d. after oral administration.

Dose proportionality of  $AUC_{\tau, ss}$  of selexipag and ACT-333679 after i.v. selexipag will be analyzed using the power model approach [Gough 1995], if at least three different dose levels with a sufficient number of subjects to compute CIs are included in the PKS. A plot of log dose versus log  $AUC_{\tau, ss}$  including the slope of the estimated parameter will be displayed.

Differences in t<sub>max, ss</sub> of ACT-333679 between the i.v. selexipag period and the Uptravi period will be assessed within each dose level using a Wilcoxon signed rank test and displaying the median estimate and exact 90% CI of the location shift using Hodges-Lehmann estimation.

If considered appropriate, a sensitivity analysis may be conducted to evaluate the statistical impact of the plasma concentrations of selexipag or ACT-333679 that were considered implausible by the PK expert.
## 8 GENERAL STATISTICAL METHODOLOGY

All analyses described in this document will be performed by the contract research organization Datamap GmbH, Freiburg, Germany using Statistical Analysis Software (SAS®) version 9.3 or higher.

## 8.1 General rules for data presentations

This section describes the general rules applied for all data displays, unless otherwise specified in each corresponding section.

Data listings will show all assessments included in the study database, regardless if used in specific summary tables.

#### 8.1.1 Summary statistics of non-PK data

Clinical data will be listed and summarized using appropriate descriptive statistics:

- For continuous variables: Number of non-missing observations, mean, standard deviation, minimum, median, and maximum.
- For dichotomous or categorical variables: Number of non-missing observations, and frequency with percentage per category. Denominators for percentages are the number of subjects in the pertinent analysis set and period, unless otherwise specified.

#### 8.1.2 Summary statistics of PK data

PK data will be listed as described in Section 7.8.4 and summarized using appropriate descriptive statistics:

- Plasma concentrations of selexipag and ACT-333679 will be summarized using number of non-missing observations, arithmetic mean, geometric mean, standard deviation (SD), standard error of the mean (SE), minimum, median, maximum and 95% CIs for the arithmetic and geometric mean.
- C<sub>trough, ss</sub> of selexipag and ACT-333679 will be summarized using number of non-missing observations, arithmetic mean, geometric mean, SD, SE, coefficient of variation of the observed and logarithmized data (CV, CV<sub>ln</sub>) in %, minimum, median, maximum and 95% CIs for the arithmetic and geometric mean.
- $C_{max, ss}$  and  $AUC_{\tau, ss}$  of selexipag and ACT-333679 will be summarized using number of non-missing observations, arithmetic mean, geometric mean, SD, SE, CV%,  $CV_{ln}$ %, minimum, median, maximum, 95% CIs for the arithmetic and geometric mean.
- t<sub>max, ss</sub> of selexipag and ACT-333679 will be summarized using number of non-missing observations, arithmetic mean, SD, SE, CV%, minimum, median, maximum and 95% CI for the arithmetic mean.

#### 8.2 Statistical methods

This section describes in general terms the statistical models and methods applied.

No confirmatory hypothesis testing will be conducted in this study. All tests and CIs will be of descriptive nature. Confidence levels are chosen as 90% for PK geometric means and 95% for all other confidence levels and will not be adapted for multiplicity.

 $C_{trough, ss}$ ,  $C_{max, ss}$ , and  $AUC_{\tau, ss}$ , values are assumed to be log-normally distributed.

#### 8.2.1 Statistical methods for discrete data

### 8.2.1.1 Exact Pearson-Clopper CIs for the incidence of AEs

Due to the small number of subjects included in the trial, broader estimates for the incidence rates of AEs need to be computed. The Pearson-Clopper method yields exact, while conservative confidence limits, i.e., the CI is at least 95%. They will be computed using PROC FREQ as shown below, assuming the input dataset contains counts for each *aedecod*, with 0 indicating subjects without event and 1 indicating subjects with event.

```
PROC FREQ data=<input_dataset>;

BY aedecod;

TABLES event /exact binomial (level='1');

WEIGHT count;

RUN;
```

#### 8.2.2 Statistical methods for continuous data

## 8.2.2.1 Differences between periods in $C_{max, ss}$ and $AUC_{\tau, ss}$ of selexipag/ACT-333679

Within each dose level and after dose normalization, differences between the Uptravi and i.v. selexipag periods will be analyzed by computing the geometric mean ratios of the respective period with the oral formulation as reference treatment in the denominator. This is done by fitting a mixed linear model to the log-transformed  $C_{max,\ ss}$  and  $AUC_{\tau,\ ss}$  values with period as fixed and subject as random effect. The Kenward-Rodgers method for calculation of degrees of freedom will be used to obtain degrees of freedom to calculate CIs. An unstructured covariance matrix will be assumed. The difference of the least squares mean and its 90% CI will be computed and transformed back to normal scale to obtain the geometric mean ratio. SAS® code similar to the code shown below will be used:

PROC MIXED data=<input\_dataset>;

CLASS period;

MODEL log\_response=period / DDFM=KR;

RANDOM intercept /subject=usubjid TYPE=UN;

ESTIMATE 'Difference i.v. - oral' period -1 1 /CL ALPHA=0.1;

RUN;

## 8.2.2.2 $CV_b$ in $C_{max, ss}$ and $AUC_{\tau, ss}$ of selexipag/ACT-333679

The CV<sub>b</sub> expressed in percent will be computed using the formula

$$CV_b [\%] = 100\sqrt{e^{S_b^2} - 1}$$

where  $S_b^2$  is the MSE of the residuals from the mixed effects model described in Section 8.2.2.1.

## 8.2.2.3 Dose proportionality of $AUC_{\tau, ss}$ of selexipag/ACT-333679

To assess dose proportionality of selexipag the power model approach will be used:

The power model approach specifies a relationship between the scheduled dose D of i.v. selexipag and  $AUC_{\tau, ss}$  of selexipag / ACT-333679 which is expressed as

$$Y_{ij} = \alpha_i$$
 \*  $D_i^{\beta}$  \*  $\epsilon'_{ij}$ 

Together with  $\alpha'$  denoting  $\exp(\alpha)$  and  $\epsilon'_{ij}$  denoting  $\exp(\epsilon'_{ij})$ , logarithmizing both sides of the equation yields a linear model

$$log(Y_{ij}) = \alpha_j + \beta log(D_i) + \epsilon_{ij}$$

with

 $Y_{ij}$  AUC<sub> $\tau$ , ss</sub> of dose level i in subject j (i=1, ..., I), (j=1, ..., n)

α<sub>i</sub> intercept parameter (assumed to be a random effect)

 $\beta$  the slope parameter

D<sub>i</sub> size of dose level i

 $\varepsilon_{ij}$  random error term of subject j in dose level i.

This model equation can be fitted using a mixed linear model with  $log(D_i)$  as a covariate and subject as random effect. The 90% CI for the parameter estimate for the covariate will be computed. In case of dose proportionality, 1 should be included in the 90% CI of the parameter estimate.

SAS® code similar to the following will be used:

```
PROC MIXED data=<input_dataset>;

MODEL log_response=log_dose / DDFM=KR S CL ALPHA=0.1;

RANDOM intercept /subject=usubjid TYPE=UN;

RUN;
```

The assessment of dose proportionality using the power approach will only be conducted when at least three dose levels are included into the study.

## 8.2.2.4 Difference of t<sub>max</sub>, ss of ACT-333679

Within each dose level, difference in  $t_{max, ss}$  of ACT-333679 between Periods 1 and 2 will be assessed by computing the Hodges-Lehmann estimator for shift in the median from Uptravi to i.v. selexipag. The median is computed by computing all shifts between the two periods and using the median of the shifts as an estimate. If computationally feasible, exact estimates and 90% CIs will be computed.

#### 9 INTERIM ANALYSIS

No interim analysis is planned in this trial.

#### 10 GENERAL DEFINITIONS AND DERIVATIONS

This section describes all recurrent general definitions (e.g., study treatment start date, baseline, study day) which will be used for the derivations of variables and summary tables and are not covered in the sections above.

### 10.1 Handling of screening and re-screening data

Data of re-screened subjects obtained at the re-screening visit will be used as 'Screening' data. If a data point is not collected at re-screening but was collected at the previous screening visit, the data point from the screening visit will be used.

## 10.2 Analysis periods and visit windows

## 10.2.1 Study treatment start and end date

The date and time of the first infusion of i.v. selexipag will be considered study treatment start date/time. The end date and time of the last infusion of i.v. selexipag will be considered study treatment end date/time.

#### 10.2.2 Study days

The day of intake of the Uptravi during pre-treatment period, i.e., Period 1 [see Section 2.3] will be considered Day 1. There is no Day 0; the day before Day 1 will be considered Day -1.

Note that study treatment will be administered on Day 2 and Day 3 according to this definition; thus study day definition corresponds to the study days used in the study protocol.

#### 10.2.3 Baseline

All assessments on Day 1 will be considered baseline. If a Day 1 assessment is not available, the last assessment prior to Day 1 will be considered baseline.

#### 10.2.4 Unscheduled visits and visit windows

Assessments made on both, scheduled and unscheduled visits will be assigned to an analysis period according to Table 2 using the assessment date and time.

Furthermore, each assessment will be assigned an analysis visit using the time windows described in Table 13. If more than one assessment was made within a visit time window, the closest value to the target Visit is displayed in by visit displays.

Table 13 Analysis visit windows

| Analysis<br>visit | Nominal<br>study day* | Lower bound<br>study day* | Upper bound study day* |
|---|---|---|---|
| Visit 2, Day 1 | Day 1 | Day of informed consent | Day 1 |
| Visit 2, Day 2 | Day 2 | Day 2 | Day 2 |
| Visit 2, Day 3 | Day 3 | Day 3 | Day 3 |
| Visit 3 | Day 12 | Day 4 | Day 22 |
| Visit 4 | Day 33 | Day 23 | End of Study |
| * Study days are defined as in Section 10.2.2. | | | |

<sup>10.3</sup> Uptravi dosage subgroups

Enrollment is controlled by an interactive response technology system based on the subject's stable Uptravi dose. For analysis purposes, the information entered into the system will determine the allocation to one of the two dosage subgroups.

## 10.4 Derived and computed variables for analysis datasets

CDISC ADaM version 2.1 and ADaM implementation guide 1.1 will be followed.

For details on the derivation of specific analysis variables, please refer to the programming specifications document.

#### 10.5 Handling of missing/incomplete date and time fields

Missing parts for specific dates/times will be changed into acceptable non-missing values as described in the table below.

| Type of date/time | Imputation method when date/time is incomplete | Imputation method when date/time is missing |
|---|---|---|
| Start Date/Time of Adverse Event | If the end date of the AE is not before the start of study treatment, and if the study treatment start falls in the range of possible dates, the study treatment start date is used. In all the other cases, the lower limit (i.e., first day of the month, 00:00h) is used. | Date & time of first i.v. selexipag |
| End Date/Time<br>of Adverse<br>Event | Use the upper limit of the range of possible dates given the nonmissing date/time parts, i.e., last day of the month or last day of the year, 23:59h | |

| Start Date of<br>Medication | If the date of the Screening visit is within the range of possible dates, use the Screening visit date. Otherwise, use first day of the month and/or first day of the year. | Date of Screening visit |
|---|---|---|
| End Date of<br>Medication | Use the upper limit of the range of possible dates given the nonmissing date/time parts, i.e., last day of the month or last day of the year | •• |
| Date of initial<br>diagnosis of<br>PAH | Day missing: 15th of the month Day and month missing: 30th of June If the resulting date is later than the date of screening visit date and the lower limit is not later than the screening visit date, then the date is substituted with the date of screening visit. | No replacement |
| PK sample<br>Date/Time | If the scheduled time is within the possible range given the nonmissing date/time parts, use the scheduled date/time. Otherwise, the sample date/time cannot be imputed. | No replacement |

## 10.6 Handling of missing infusion durations

If the start time or end time of the infusion or the time point of the infusion rate increase is missing, study treatment administration times as stipulated in the protocol will be assumed for analysis, i.e., 15 min duration of the initial infusion rate and 72 min of the increased infusion rate.

## 11 CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL

This section describes changes to the statistical analysis planned in the protocol, and other deviations from the protocol relevant to the analysis or interpretation of the results.

## 11.1 Changes to the analyses planned in the study protocol None.

## 11.2 Changes in the conduct of the study / data collection None.

# 11.3 Clarifications concerning endpoint definitions and related variables or statistical methods

#### 11.3.1 Treatment/period as factor in mixed model analysis

Protocol section 10.3.5 [D-17.055] states that the mixed model analysis of  $C_{max, ss}$  and  $AUC_{\tau, ss}$  contains terms for period, treatment and subject. Since 'period' and 'treatment' are confounded (Period 1: Uptravi, Period 2: i.v. Selexipag) only 'period' is used in the models.

### 11.3.2 Additional analyses as compared to the study protocol

- C<sub>trough</sub> ratio of treatments per subject.
- Marked blood pressure abnormalities.

### 12 LIST OF TABLES, LISTINGS AND FIGURES

Since all tables, figures, and listings will be produced using SAS®, the outputs actually generated may slightly differ from the mock-ups presented in the study-specific mock-up catalogue.

## 12.1 Subject disposition

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| DISP | T | Subject disposition | SCR | Y | T_DISP |
| DISP_COU | T | Subject disposition by country and site | SCR | | T DISP CO<br>U |
| ANA | T | Overview of analysis sets and reasons for exclusion from analysis sets | SCR | | T_ANA |
| PWDS | T | Reasons for premature discontinuation from the study | SAF | | T_PWDS |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

#### 12.2 Protocol deviations

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| PD | T | Summary of important protocol deviations | SCR | | T_PD |
| PD_COU | T | Summary of all protocol deviations overall and by country | SCR | | T_PD |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.3 Subject characteristics

## 12.3.1 Demographics and baseline disease characteristics

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| DEM | T | Summary of baseline demographic characteristics | SAF | Y | T_DEM |
| AGECATE<br>U | Т | EudraCT age categories | SAF | | T_AGECATE<br>U |
| BAS | T | Summary of baseline disease characteristics | SAF | Y | T_BAS |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF=i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

#### 12.3.2 Other baseline characteristics

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| PHYS | L | Listing of physical examination results | SCR | | L_PHYS |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

### 12.3.3 Medical history

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| MH_PRV_<br>SOC | T | Summary of previous diseases or<br>diagnoses, by primary system organ<br>class and preferred term | SAF | | T_MH_SOC |
| MH_ONG_<br>SOC | T | Summary of concomitant diseases or diagnoses, by primary system organ class and preferred term | SAF | | T_MH_SOC |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF=i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.3.4 Previous and concomitant medications

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| CM_PRV | T | Summary of previous therapies by Anatomical Therapeutic Chemistry (ATC) Class and Preferred Term [Add footnote: Previous therapies are therapies which ended prior to baseline.] | SAF | | T_CM |
| CM_ONG | T | Summary of ongoing therapies by Anatomical Therapeutic Chemistry (ATC) Class and Preferred Term [Add footnote: Ongoing therapies are therapies which were started prior to baseline and are ongoing at study treatment start.] | SAF | | T_CM |
| CM_CM | T | Summary of study concomitant therapies by Anatomical Therapeutic Chemistry (ATC) Class and Preferred Term [Add footnote: Study concomitant therapies are therapies which were started or dose changed (of those ongoing at baseline) during the respective period.] | SAF | | T_CM |
| CM_ONG_<br>PAH | T | Summary of ongoing PAH specific therapies at baseline [Add footnote: Ongoing therapies at study treatment start are therapies which were started prior to baseline and are ongoing at study treatment start.] | SAF | Y | T_CMPAH |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.4 Study treatment exposure

#### 12.4.1 Exposure

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| EXP_IV | T | Exposure to i.v. selexipag | ivSAF | Y | T_EXP_IV |
| EXP_PO | T | Exposure to Uptravi prior to and after i.v. selexipag | SAF<br>ivSAF# | | T_EXP_PO |
| COMPL_I<br>V | T | Compliance to study treatment | ivSAF | | T_COMPL_I<br>V |
| EXP_ADJ | T | Summary of study treatment administration, reasons for interruptions and end of infusion | ivSAF | | T_EXP_ADJ |
| EXP_SHF | F | Shift in selexipag dose between oral and i.v. treatment | ivSAF | | F_EXP |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

## 12.4.2 Study treatment discontinuation

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| PWDT | T | Reasons for premature discontinuation of i.v. selexipag treatment | ivSAF | | T_PWDT |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF=i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.5 Study withdrawal

See Section 12.4.

## 12.6 Primary efficacy analyses

Not applicable.

## 12.7 Safety analyses

#### 12.7.1 Adverse events

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| AE_ALL_S<br>OC | T | Incidence of adverse events by period,<br>primary system organ class and<br>preferred term | | Y | T_AE_SOC |
| AE_INT | T | Incidence of adverse events by preferred term and maximum intensity | SAF<br>ivSAF# | | T_AE_PT_IN<br>T |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

#### 12.7.2 Deaths and serious adverse events

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| SAE_ALL_<br>PT | T | Incidence of serious adverse events by period, and preferred term | SAF<br>ivSAF# | Y | T_AE_PT |
| DTH | L | Listing of all deaths | SAF | | L_DTH |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

### 12.7.3 Prostacyclin-associated adverse events

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_PC_PT | T | Incidence of prostacyclin-associated adverse events by period and preferred term | | Y | T_AE_PT |
| SAE_PC_P<br>T | T | Incidence of prostacyclin-associated serious adverse events by period and preferred term | | | T_AE_PT |
| AE_PCDC<br>_PT | T | Incidence of prostacyclin-associated<br>adverse events leading to<br>discontinuation of study treatment by<br>preferred term | | | T_AE_PT |

## 12.7.4 Adverse events of special interest based on the Uptravi risk management plan

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_RMP | T | Incidence of adverse events of special interest based on the Uptravi risk management plan by period, risk category and preferred term [Replace SOC with Risk category in the Shell Delete SOC on footnote regarding MedDRA version] | SAF<br>ivSAF# | | T_AE_SOC |
| SAE_RMP | L | Listing of all serious adverse events of special interest based on the Uptravi risk management plan [Replace SOC with Risk category in the Shell.] | SAF<br>ivSAF# | | L_AE |
| AE_DC_R<br>MP | T | Incidence of adverse events of special interest based on the Uptravi risk management plan leading to discontinuation of study treatment by period, risk category and preferred term [Replace SOC with Risk category in the Shell. Delete SOC on footnote regarding MedDRA version.] | SAF<br>ivSAF# | | T_AE_SOC |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

## 12.7.5 Injection site reaction adverse events

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_INJ_IN<br>T | T | Incidence of clinically significant injection site reaction adverse events by preferred term and maximum intensity | ivSAF | Y | T_AE_PT_IN<br>T |
| AE_INJDE<br>T | T | Grade and diagnosis criteria of injection site reactions | ivSAF | | T_AEINJ |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF=i.v. Safety analysis set, PKS=Pharmacokinetic analysis set.

#### 12.7.6 PAH-related adverse events

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_PAH_<br>PT | Т | Incidence of PAH related adverse events by period and by preferred term | SAF<br>ivSAF# | | T_AE_PT |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

#### 12.7.7 Adverse events leading to study treatment discontinuation

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_DC_P<br>T | T | Adverse events leading to discontinuation of study treatment by preferred term | ivSAF | | T_AE_PT |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set.

## 12.7.8 Adverse events related to study drug

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| AE_REL_P<br>T | T | Incidence of adverse events related to<br>study treatment as judged by the<br>investigator by period and by preferred<br>term | ivSAF | | T_AE_PT |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set.

## 12.7.9 Summaries of adverse events for disclosure

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliv<br>erabl<br>e | Mock layout |
|---|---|---|---|---|---|
| SAE_CTG<br>OV | T | Summary of treatment emergent SAEs | SAF | | T_AE_SOC2 |
| SAE_REL_<br>CTGOV | T | Summary of treatment emergent SAEs judged to be treatment related by the investigator | SAF | | T_AE_SOC2 |
| SAE_DTH<br>_CTGOV | T | Summary of treatment emergent SAEs with fatal outcome | SAF | | T_AE_SOC2 |
| SAE_DTH<br>REL_CTG<br>OV | T | Summary of treatment emergent SAEs with fatal outcome judged to be treatment related by the investigator | SAF | | T_AE_SOC2 |
| NSAE_5PC<br>T_CTGOV | T | Summary of non-serious AEs with an incidence of 5% or higher in any treatment group | SAF | | T_AE_SOC2 |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.7.10Laboratory tests

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| LB_SUM_<br>HEM | T | Summary and change from baseline of hematology values, by visit | SAF<br>ivSAF# | | T_LB_SUM |
| LB_SUM_<br>CHE | T | Summary and change from baseline of biochemistry values, by visit | SAF<br>ivSAF# | | T_LB_SUM |
| LB_ABN_<br>P2 | T | Incidence of marked laboratory values, by period | SAF<br>ivSAF# | | T_LB_ABN |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

## 12.7.11Vital signs and body weight

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliverab<br>le | Mock<br>layout |
|---|---|---|---|---|---|
| VS_WGT_<br>SUM | T | Summary and change from baseline of body weight, by visit | SAF<br>ivSAF# | | T_LB_SU<br>M |
| VS_SUM | T | Summary and change from baseline of vital signs, by visit | SAF<br>ivSAF# | | T_VS_SU<br>M |
| VS_PRED<br>S | T | Summary of post-dose values and change from pre-dose of vital signs, by visit | | Y | T_VS_PR<br>EDS |
| VS_ABN | T | Incidence of marked blood pressure abnormalities, by period | SAF<br>ivSAF# | Y | T_VS_A<br>BN |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

#### 12.7.12ECG

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock<br>layout |
|---|---|---|---|---|---|
| EG_SUM | T | Summary and change from baseline of quantitative ECG parameters, by visit | SAF<br>ivSAF# | | T_EG_SU<br>M |
| EG_PRED | T | Summary of post-dose values and change from pre-dose of quantitative ECG parameters, by visit | | | T_EG_PRE<br>DS |
| EG_QUAL<br>_SUM | T | Summary of qualitative ECG findings, by visit | SAF<br>ivSAF# | | T_EG_QU<br>AL |
| EG_ABN | T | Incidence of ECG abnormalities - QT prolongation, by period | SAF<br>ivSAF# | | T_EG_AB<br>N |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

## 12.7.13WHO Functional class

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| WHO_SU<br>M | T | Summary of WHO functional class, by visit [include a best/worst post baseline category] | SAF<br>ivSAF# | | T_WHO_SU<br>M |
| WHO_CH<br>G | T | Shift table of WHO functional class from baseline to each study visit [include a shift to worst/best post baseline category] | | | T_WHO_CH<br>G |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set, # Tables will run on SAF only if SAF and ivSAF are identical.

## 12.8 PK analyses

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| PK_CON_<br>SUM_SEL | T | Summary of selexipag plasma concentrations [ng/mL] per time point by dose level and treatment | PKS | | T_PK_CON_<br>SUM |

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| PK_CON_<br>SUM_ACT | T | Summary of ACT-333679 plasma concentrations [ng/mL] per time point by dose level and treatment | PKS | | T_PK_CON_<br>SUM |
| PK_EP_SU<br>M_SEL | T | Summary of PK endpoints of selexipag by dose level and treatment | PKS | Y | T_PK_EP_S<br>UM |
| PK_EP_SU<br>M_ACT | T | Summary of PK endpoints of ACT-333679 by dose level and treatment | PKS | Y | T_PK_EP_S<br>UM |
| PK_SUM_<br>RATIO | T | Summary of PK parameters of ratio ACT-333679/selexipag concentration by dose level and treatment | PKS | | T_PK_RATI<br>O_SUM |
| PK_MM_S<br>EL | T | Mixed model analysis: Ratio of Uptravi<br>and i.v. selexipag period for selexipag<br>by dose level | PKS | Y | T_PK_MM |
| PK_MM_A<br>CT | T | Mixed model analysis: Ratio of Uptravi<br>and i.v. selexipag period for ACT-<br>333679 by dose level | PKS | Y | T_PK_MM |
| PK_POW_<br>AUC_SEL | T | Dose proportionality of AUCtau of selexipag after i.v. selexipag: Power model estimation | PKS | Y | T_PK_POW |
| PK_POW_<br>AUC_SEL | F | Dose proportionality of AUCtau of selexipag after i.v. selexipag: Power model estimation | PKS | Y | F_PK_POW |
| PK_POW_<br>AUC_ACT | T | Dose proportionality of AUCtau of ACT-333679 after i.v. selexipag: Power model estimation | PKS | Y | T_PK_POW |
| PK_POW_<br>AUC_ACT | F | Dose proportionality of AUCtau of ACT-333679 after i.v. selexipag: Power model estimation | PKS | Y | F_PK_POW |
| PK_WIL_S<br>EL | T | Location shift analysis of tmax, ss of selexipag | PKS | | T_PK_WIL |
| PK WIL<br>ACT | T | Location shift analysis of tmax, ss of ACT-333679 | PKS | | T_PK_WIL |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

## 12.9 Subject listings

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| SCRF | L | Listing of screening failures | SCR | | L_SCRF |
| PWDS | L | Listing of reasons for premature discontinuation from the study | SAF | | L_PWDS |
| PD | L | Listing of protocol deviations | SCR | | L_PD |
| ANSET | L | Listing of analysis sets | SCR | | L_ANSET |
| PWDT | L | Listing of reasons for premature discontinuation of i.v. selexipag treatment | ivSAF | | L_PWDT |
| DEM | L | Listing of demographics | SCR | | L_DEM |
| BAS | L | Listing of baseline disease characteristics | SCR | | L_BAS |
| MH | L | Listing of medical history | SAF | | L_MH |
| CM | L | Listing of previous and concomitant therapies | SAF | | L_CM |
| CM_PAH_<br>MOD | L | Listing of PAH specific therapies newly started dose changed or stopped during any period. [Add footnote: Interruptions of Uptravi during i.v. selexipag period as mandated in the protocol are not shown.] | SAF | | L_CM |
| EXP_PO | L | Listing of Uptravi dosing records | SAF | | L_EXP_PO |
| EXP_IV | L | Listing of study treatment dosing records | ivSAF | | L_EXP_IV |
| COMP | L | Listing of compliance | ivSAF | | L_COMP |
| AE | L | Listing of all adverse events | SCR | | L_AE |
| AE_SCR | L | Adverse events in the Screening Period prior to the first dose of Uptravi on Visit 2 Day 1 | SCR | | L_AE |
| AE_DTH | L | Listing of all adverse events leading to death | SAF | | L_AE |
| SAE | L | Listing of all serious adverse events | SAF | | L_AE |

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Key<br>deliver<br>able | Mock layout |
|---|---|---|---|---|---|
| AE_PC | L | Listing of all prostacyclin-associated adverse events | SAF | | L_AE |
| AE_RMP | L | Listing of all adverse events of special interest based on the Uptravi risk management plan [Replace SOC with Risk category in the Shell. Delete SOC on footnote regarding MedDRA version.] | SAF | | L_AE |
| AE_INJDE<br>T | L | Listing of all injection site reactions | ivSAF | | L_AEINJ |
| AE_PAH | L | Listing of PAH related adverse events | SAF | | L_AE |
| AE_DC | L | Listing of adverse events leading to discontinuation of study treatment | ivSAF | | L_AE |
| AE_REL | L | Listing of adverse events related to<br>study treatment as judged by the<br>investigator | ivSAF | | L_AE |
| LAB | L | Listing of laboratory parameters | SCR | | L_LAB |
| VS | L | Listing of vital signs, body weight and height | SCR | | L_VS |
| EG | L | Listing of quantitative ECG measurements | SAF | | L_EG |
| EG_QUAL | L | Listing of qualitative ECG findings | SAF | | L_EG_QUAL |
| WHO | L | Listing of WHO functional class | SCR | | L_WHO |
| PK_CONC | L | Listing of selexipag / ACT-333679 plasma concentrations | PKS | | L_PK_CONC |
| PK_DER | L | Listing of derived PK parameters of selexipag and ACT-333679 | PKS | | L_PK_DER |
| PK_RATIO | L | Listing of Cmax,ss and AUCtau,ss ratio of ACT-333679/selexipag | PKS | | L_PK_RATI<br>O |
| IMP_CON<br>C | L | Listing of selexipag concentration in the infusion solution | PKS | | L_IMP_CON<br>C |

<sup>\*</sup> T=Summary table, L=Listing, F=Figure, \*\*SCR=Screened analysis set, SAF=Safety analysis set, ivSAF= i.v. Safety analysis set, PKS=Pharmacokinetic analysis set

#### 13 REFERENCES

[D-17.055] AC-065A309: A multicenter, open-label, single-sequence crossover study to assess safety, tolerability and pharmacokinetic of intravenous selexipag in subjects with stable pulmonary arterial hypertension transitioning from an oral stable dose of selexipag. Clinical Study Protocol Version 1. Actelion Pharmaceuticals Ltd; 27 January 2017.


[Gough 1995] Gough K, Hutchinson M, Keene O, Byrom B, Ellis S, Lacey L, et al Assessment of dose proportionality: Report from the statisticians in The Pharmaceutical Industry/Pharmacokinetics UK joint working party. Drug Information Journal. 1995;29:1039–48.

## 14 APPENDICES

## Appendix A Protocol synopsis

## PROTOCOL SYNOPSIS AC-065A309

| TITLE | A multicenter, open-label, single-sequence cross-over study to |
|---|---|
| | assess safety, tolerability, and pharmacokinetics of intravenous |
| | selexipag in subjects with stable pulmonary arterial hypertension |
| OBJECTIVES | switching from an oral stable dose of selexipag Primary objective(s) |
| OBJECTIVES | The primary objective of this study is to assess whether temporary |
| | switching from a stable oral dose of selexipag to an intravenous |
| | (i.v.) dose of selexipag providing comparable exposure to active |
| | metabolite ACT-333679 and switching back to the initial oral |
| | dose of selexipag is safe and well tolerated in subjects with stable pulmonary arterial hypertension (PAH). |
| | Other objectives |
| | Other objectives are described in Section 2.2. |
| DESIGN | This is a prospective, multi-center, open-label, single-sequence, |
| | cross-over, Phase 3 study. |
| | Subjects with stable PAH, currently treated with Uptravi® at a |
| | stable dose (i.e., unchanged dose for 28 days), will be enrolled. |
| | Subjects will be hospitalized during Period 1 (pre-treatment |
| | period) and Period 2 (treatment period). |
| | No interim analysis is planned. |
| PERIODS | Screening period: |
| | Up to 28 days; starts with the signing of the Informed Consent |
| | Form (ICF) and ends with first day (Visit 2, Day 1) of Period 1 |
| | (Uptravi, pre-treatment period). |
| | Treatment and observation period: |
| | The treatment and observation period includes the following |
| | consecutive periods: |
| | • Period 1 (Uptravi, pre-treatment period, in-hospital): 1 day |
| | Starts with intake of the morning dose of Uptravi at Visit 2 Day |
| | 1 and ends the following day, before initiation of the first |
| | infusion of i.v. selexipag. |
| | • Period 2 (i.v. selexipag, treatment period, in-hospital): 36 hours |
| | (3 doses) Starts in the marning of Visit 2 on Day 2 with the start of the |
| | Starts in the morning of Visit 2 on Day 2 with the start of the |

| | first infusion of i.v. selexipag and ends in the evening of Visit 2 |
|---|---|
| | <ul> <li>on Day 3 before the evening administration of Uptravi. Note: oral administration of Uptravi is interrupted during the treatment period with i.v. selexipag.</li> <li>Period 3 (Uptravi, post-treatment period): 7 to 11 days Starts in the evening of Visit 2 on Day 3 with the oral administration of Uptravi and ends 7 to 11 days later, at Visit 3.</li> <li>Safety Follow-up period: Starts at the end of Visit 3 and ends 30 to 37 days after the last administration of i.v. selexipag with the End-of-Study telephone call (Visit 4).</li> </ul> |
| PLANNED<br>DURATION | Approximately 9–12 months from first subject first visit to last subject last visit. |
| SITE(S) /<br>COUNTRY(IES) | 10 sites in 2 countries (planned). |
| SUBJECTS /<br>GROUPS | <ul> <li>Approximately 20 subjects will be enrolled in order to obtain 18 evaluable subjects.</li> <li>Two different groups of subjects will be enrolled based on their dose of Uptravi:</li> <li>Group A: Subjects with a stable dose of Uptravi between 200 and 1000 μg twice daily (b.i.d.; inclusive): at least 5 and up to 8 subjects will be enrolled in this dose group.</li> <li>Group B: Subjects with a stable dose of Uptravi between</li> </ul> |
| | 1200 and 1600 μg b.i.d. (inclusive): At least 12 and up to 15 subjects will be enrolled in this dose group. |
| INCLUSION<br>CRITERIA | <ol> <li>Signed ICF prior to any study-mandated procedure.</li> <li>Male and female subjects at least 18 to 75 years inclusive.</li> <li>Subjects with PAH belonging to the Updated Clinical Classification Group 1 [Galiè 2016]</li> <li>Subjects who have been prescribed Uptravi in compliance with local prescribing information (i.e., SmPC or USPI).</li> <li>Stable PAH defined as WHO Functional Class (FC) I–III at Visit 1 and Visit 2 and no change (i.e., introduction or dose change) in PAH-specific medication (i.e., ERA, PDE-5 inhibitor or sGC stimulator) and diuretics in the last 28 days prior to Visit 2.</li> <li>Subjects currently treated with Uptravi at a stable dose (i.e., unchanged dose) for at least 28 days before Visit 2.</li> <li>A woman of childbearing potential is eligible only if she has a negative urine pregnancy test at Visit 1 and at Visit 2.</li> </ol> |
| EXCLUSION | 1. Pregnant, planning to become pregnant or lactating. |

| CRITERIA | 2. Known and documented moderate or severe hepatic impairment. |
|---|---|
| | 3. Subjects having received gemfibrozil at any time since |
| | initiation of Uptravi. |
| | 4. Treatment with any prostacyclin and prostacyclin analogs |
| | within 28 days prior to Visit 1. 5. SBP < 90 mmHg at Visit 1 or at Visit 2. |
| | 6. Known or suspected uncontrolled hyperthyroidism. |
| | 7. Severe renal failure and ongoing or planned dialysis. |
| | 8. Any known factor or disease that might interfere with |
| | treatment compliance, study conduct, or interpretation of the |
| | results, such as drug or alcohol dependence or psychiatric |
| | disease. |
| | 9. Known concomitant life-threatening disease with a life expectancy < 12 months. |
| | 10. Treatment with another investigational treatment within 3 months of Visit 1. |
| STUDY | Investigational treatment |
| TREATMENTS | The study treatment (i.v. selexipag) will be administered b.i.d. intravenously as an infusion over an 87 minute period [see Section 5.1.4]. The dose of i.v. selexipag will be individualized for each subject and will aim to reach an exposure to the active metabolite (area under the concentration-time curve [AUC] between two doses) comparable to the one obtained with subject's current oral dose of Uptravi. |
| | Comparator and/or placebo<br>Not applicable. |
| AUXILIARY<br>MEDICINAL<br>PRODUCTS | The study population consists of subjects who have been prescribed Uptravi (oral selexipag) as part of their standard PAH treatment (i.e., Uptravi must not have been prescribed solely for the purpose of the study). Subjects will keep using Uptravi during their participation in the study as prescribed by their physician and in compliance with the USPI/SmPC [Uptravi® SmPC; Uptravi® USPI] including the use of contraception for women of childbearing potential. Subject's oral treatment with Uptravi will be temporarily interrupted for 36 hours during the administration of study treatment (i.v. selexipag). |
| ENDPOINTS | Primary efficacy endpoint(s) |
| | Not applicable. |
| | Secondary efficacy endpoints Not applicable. |

| | 7 |
|---|---|
| | Main safety and tolerability endpoints The main safety and tolerability endpoints will be analyzed over the Period 1, Period 2, and Period 3 combined. |
| | - Discontinuations due to prostacyclin-associated adverse events (AEs). |
| | - AEs and serious AEs (SAEs). |
| | - Prostacyclin-associated AEs. |
| | - AEs related to injection site reactions. |
| | - PAH-related AEs. |
| | Other endpoints |
| | Other endpoints are described in Section 6.2.3. |
| PHARMACOKINETIC ENDPOINTS | ( 1, 33) |
| L. I.D. G. III. G | selexipag and its active metabolite, ACT-333679, at steady state after Uptravi (oral selexipag) in Period 1 and after i.v. |
| | selexipag administration in Period 2. |
| | - The maximum plasma concentration at steady state $(C_{max, ss})$ of |
| | selexipag and its active metabolite, ACT-333679 after Uptravi |
| | (oral selexipag) in Period 1 and i.v. selexipag administration in |
| | Period 2. - The time to reach maximum plasma concentration at steady-state |
| | The time to reach maximum plasma concentration at steady-state $(t_{\text{max, ss}})$ of selexipag and its active metabolite, ACT-333679 after |
| | Uptravi (oral selexipag) in Period 1 and i.v. selexipag |
| | administration in Period 2. |
| | • Trough plasma concentration at steady state (C <sub>trough, ss</sub> ) of |
| | selexipag and its active metabolite, ACT-333679after Uptravi (oral selexipag) in Period 1 and i.v. selexipag administration in Period 2. |
| ASSESSMENTS | Refer to the schedule of assessments in Table 2. |
| STATISTICAL | Approximately 20 patients will be enrolled. In the GRIPHON |
| METHODOLOGY | Phase 3 pivotal study of selexipag, a proportion of 7.5% of |
| | patients on selexipag prematurely discontinued the study (i.e., |
| | without a morbidity/mortality event) due to prostacyclin-<br>associated AEs. It is expected that the proportion of |
| | discontinuations will not be higher than 10%. |
| | The statistical analysis will be mainly descriptive, i.e., no hypotheses will be formally tested. |
| | Four analysis sets are defined in this study: |
| | - Screened Analysis Set includes all subjects who are screened and have a subject identification number. |

- i.v. Safety Set comprises all subjects who received at least one dose of i.v. study treatment.
- Safety Set (SAF) includes all enrolled (included in the study on Day 1) subjects who receive at least one dose of selexipag (oral or i.v.).
- Pharmacokinetic Analysis Set (PKS) comprises all subjects included in the SAF who received the 3 doses of i.v. study treatment and who complied with the protocol sufficiently and did not deviate from the protocol in a way that might affect the PK outcome of the study.

The study comprises 3 main periods for analysis: Period 1, Period 2, and Period 3 and follow-up. AEs and SAEs will be tabulated, for the Safety Set and i.v. Safety Set, overall across periods as well as by study period. The proportion of discontinuations due to prostacyclin-associated AEs will be tabulated for the i.v. Safety Set and the SAF to address the primary objective. Due to the sample size, the proportion will be provided with a conservative 95% Clopper-Pearson confidence interval based on exact methods.

All secondary safety endpoints will be listed and tabulated in Safety Set and i.v. Safety Set.

Exposure will be summarized.

ECG abnormalities and laboratory variables will be descriptively summarized, both longitudinally across the study periods as well as separately per period. Death will be summarized by cause, by period, and overall.

The proportion of patients in each WHO FC (I, II, III and IV) will be tabulated at baseline and post-baseline, as well as the change in WHO FC at all assessed time points. Also the absence of worsening in WHO FC will be tabulated (i.e., patients that are either stable or improve).

## Appendix B Visit and assessment schedule

| PERIODS | Name | SCREENING | TRE | TREATMENT AND OBSERVATION PERIOD | | | | FOLLOW-UP |
|---|---|---|---|---|---|---|---|---|
| | | | Period 1 | | Period 2 | | Period 3 | |
| | | | (Pre-treatment Period; | (Treatme | nt Period; i.v. | selexipag) | (Post-treatment | |
| | | | Uptravi) | ` | | . 0, | Period; Uptravi) | |
| VISITS1 | SITS <sup>1</sup> Number Visit 1 Visit 2 | | Visit 3 | Visit 4 (Phone call) | | | | |
| | Name | Screening | Baseline | | | | | EOS |
| | Time | Day -28 to Day -1 | Day 1 | Day 2 | Day 2 | Day 3 | Day 12 (± 2days) | 30 to 37 days after |
| | | | | IV-1 (AM) | IV-2 (PM) | IV-3 (AM) | | i.v. study treatment |
| | | | | | | | | discontinuation |
| Informed co | onsent | X | | | | | | |
| Eligibility | | X | X | | | | | |
| Demographi | ics / Medical history | X | | | | | | |
| WHO FC | | X | X | | | $X^2$ | X | |
| Previous/cor | ncomitant therapy | X | X | X | X | X | X | X |
| Physical exa | mination | X | | | | | X | |
| Vital signs ( | BP, pulse rate) | X | X | X <sup>5</sup> | | X <sup>5</sup> | X | |
| Body weight | t and Height <sup>3</sup> | X | X | | | X | X | |
| Hospitalizat | ion <sup>4</sup> ** | | <del></del> | | | $\rightarrow$ | | |
| Laboratory | tests* | X | $X^6$ | | | X | X | |
| 12-lead ECC | G* | | X | $X^7$ | $X^7$ | $X^7$ | X | |
| Urine pregn | ancy test** | X | X | | | | | X |
| PK sampling | $\mathbf{g}^8$ | | X | | | X | | |
| Study treatm<br>(i.v. selex | nent administration<br>xipag) | | | X | X | X | | |
| ` | ution sampling <sup>9</sup> | | | X | X | X | | |
| SAEs/AEs <sup>10</sup> | | X | X | X | X | X | X | X |

AE = adverse event; BP = blood pressure; ECG = electrocardiogram; EOS = End-of-Study; FC = Functional Class; i.v. = intravenous; PK = pharmacokinetic; SAE = serious adverse event; WHO = World Health Organization. \*Electronically transferred to sponsor. \*\* Assessment not collected in CRF


Statistical Analysis Plan Doc No D-18.239

- 1 Unscheduled visits may be performed at any time during the study. Assessments performed during unscheduled visits are at the discretion of the investigator.
- 2 On Day 3, WHO FC is to be assessed at the end of the i.v. selexipag infusion.
- 3 Height will be assessed at Visit 1 (screening) only.
- 4 In-patient hospitalization of subjects is mandatory during Visit 2 (Period 1 and Period 2) (i.e., 2 overnight stays from Day 1 to Day 3). For convenience, the hospitalization may be extended to the night before Day 1 and to the night of Day 3.
- 5 Vital signs (BP and pulse rate) will be assessed at 7 different time points.
- 6 If Visit 1 and Visit 2 Day 1 are performed within 7 days, laboratory tests and physical examination do not have to be repeated at Visit 2 Day 1.
- 7 ECG will be performed at pre-dose and within 30 minutes after stopping of infusion (i.v. selexipag).
- 8 PK profile includes 7 blood samples.
- 9 Infusion solution samples will be taken from the tubing before each infusion.
- 10 All AEs and SAEs that occur after signing the Informed Consent Form and up to 30 days after i.v. selexipag study treatment discontinuation must be reported.

methods

Discussion and further considerations of the applied statistical

Not applicable.

**Appendix C** 

## Appendix D Definitions of marked abnormalities and elevated liver function tests

Table 14 Thresholds for marked laboratory abnormalities

| Laboratory test name | LL | LLL | нн | ННН |
|---|---|---|---|---|
| Hemoglobin (g/L) | < 100 | < 80 | Increase of > 20 g<br>above baseline | y/LIncrease of > 40 g/L<br>above baseline |
| Hematocrit (L/L) | < 0.28 (female) | < 0.20 | > 0.55 (female) | > 0.65 |
| | < 0.32 (male) | | 0.60 (male) | |
| Platelet count (10E9/L) | < 75 | < 50 | > 600 | > 999 |
| Leukocytes (10E9/L) | < 3.0 | < 2.0 | > 20.0 | > 100.0 |
| Neutrophils (10E9/L) | < 1.5 | < 1.0 | NA | NA |
| Eosinophils (10E9/L) | NA | NA | > 5.0 | NA |
| Lymphocytes (10E9/L) | < 0.8 | < 0.5 | > 4.0 | > 20 |
| ALT (U/L) | NA | NA | $> 3 \times ULN$ | > 5 × ULN |
| AST (U/L) | NA | NA | $> 3 \times ULN$ | > 5 × ULN |
| Alkaline phosphatase (U/L) | NA | NA | > 2.5 × ULN | > 5 × ULN |
| Total bilirubin (µmol/L) | NA | NA | > 2 × ULN | $> 5 \times ULN$ |
| Creatinine (µmol/L) | NA | NA | > 1.5 × ULN | $> 3 \times ULN$ |
| Sodium (mmol/L) | NA | < 130 | > 150 | > 155 |
| Potassium (mmol/L) | < 3.2 | < 3.0 | > 5.5 | > 6.0 |

ALT = alanine aminotransferase; AST = aspartate aminotransferase; NA = not applicable; SI = international system of units; ULN = upper limit of normal.

#### Appendix E Mock layout

## T DISP

ACT-293987 Protocol: AC-065A309 Subject disposition Analysis Set: Screened Analysis Set

| | Uptravi b<br>200-1000 | .i.d. dose<br>1200-1600 | |
|---|---|---|---|
| | ug<br>N=xxx<br>n (%) | ug<br>N=xxx<br>n (%) | Total<br>N=xxx<br>n (%) |
| Subjects screened<br>Screening failures | | | xxx<br>xxx |
| Subjects enrolled in Period 1<br>Subjects received Uptravi in Period 1 | xxx (100)<br>xxx (xx.x) | ( / | |
| Subjects entered in Period 2 Subjects received i.v. infusion 1 Subjects received i.v. infusion 2 Subjects received i.v. infusion 3 Subjects completed i.v. selexipag Subjects discontinued i.v. selexipag | XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| Subjects entered in Period 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects completed the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects discontinued the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Percentages are based on the number of enrolled subjects Output: <output name="">, Produced by DATAMAP on ddMMMyyyy SDTM Date: ddMMMyyyy Program: /<folder>/<pre>/<pre>program_name&gt;.sas Page x of y</pre></pre></folder></output> | | | |

Programming note: Display all categories in shell.

## T DISP COU

ACT-293987 Protocol: AC-065A309 Subject disposition by country and site Analysis Set: Screened Analysis Set

Display all categories in shell.

| Country | Uptravi b | o.i.d. dose | |
|---|---|---|---|
| Site | | 1200-1600 ug | Total |
| Periods | n (%) | n (%) | n (%) |
| Germany | | | |
| All Sites | | | |
| Subjects screened | | | XXX |
| Screening failures | | | XXX |
| Subjects enrolled in Period 1 | xxx (100) | xxx (100) | xxx (100) |
| Subjects received Uptravi in Period 1 | XXX (XX.X) | | XXX (XX.X) |
| babjeede leeelvea opelavi in leilea i | 11111 (111111) | () | () |
| Subjects entered in Period 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects received i.v. infusion 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects received i.v. infusion 2 | xxx (xx.x) | | |
| Subjects received i.v. infusion 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects completed i.v. selexipag | xxx (xx.x) | | |
| Subjects discontinued i.v. selexipag | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects entered in Period 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects completed the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects discontinued the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Site 1001 | | | |
| Subjects screened | | | XXX |
| Screening failures | | | XXX |
| Percentages are based on the number of enrolled | | | |
| Output: <output name="">, Produced by DATAMAP on dd</output> | плитадада пи:шш (сел.) | , | |
| SDTM Date: ddMMMyyyy | | | |

SDTM Date: ddMMMyyyy Program: /<folder>/<program\_name>.sas Page x of y Programming note: Include all countries and sites where subjects were enrolled.

## T ANA

ACT-293987 Protocol: AC-065A309 Overview of analysis sets and reasons for exclusion from analysis sets Analysis Set: Screened Analysis Set

| | Uptravi b.i.d. dose | | | | | |
|---|---|---|---|---|---|---|
| | | 1000 ug<br>(%) | | -1600 ug<br>(%) | | otal<br>(%) |
| Screened analysis set | | | | | ; | xxx |
| Safety analysis set | XXX | (100) | XXX | (100) | xxx | (100) |
| Subjects included in i.v. Safety analysis set | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| Subjects excluded from i.v. Safety analysis set | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 1=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 2=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 3=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| Subjects included in Pharmacokinetic analysis set | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| Subjects excluded from Pharmacokinetic analysis set | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 1=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 2=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| <reason 3=""></reason> | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| Percentages are based on the Safety analysis set Output: <output name="">, Produced by DATAMAP on ddMMMyyyy SDTM Date: ddMMMyyyy Program: /<folder>/<pre>program_name&gt;.sas Page x of y</pre></folder></output> | y hh:mm | (CET), | | | | |

Programming note: Sort reasons for exclusion in descending order of frequency. Display all categories in shell.

#### T PWDS

ACT-293987 Protocol: AC-065A309 Reasons for premature discontinuation from the study Analysis Set: Safety Analysis Set

| | Uptravi b.i.d. dose | | |
|---|---|---|---|
| | 200-Ī000 ug | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| | n (%) | n (%) | n (%) |
| Subjects completed the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects prematurely discontinued the study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lost to follow-up | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subject decision/Withdrawal of consent | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 1=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Physician decision | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <pre><reason 1=""></reason></pre> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Sponsor decision | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 1=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>//program\_name>.sasPage x of y

Programming note: Show all categories written out in the shell in the given order, even if they have zero subjects. Show reason categories as they occurred in descending frequency.

Doc No D-18.239

## $T_{-}PD$

ACT-293987 Protocol: AC-065A309 <Table title> Analysis Set: Screened Analysis Set

Overall

| | Total<br>N=xxx<br>n (%) |
|---|---|
| Subjects with at least one <important> protocol deviation</important> | xxx (xx.x) |
| <category 1=""> <deviation 1=""> <deviation 2=""> <deviation 3=""></deviation></deviation></deviation></category> | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| <category 2=""> <deviation 1=""> <deviation 2=""> <deviation 3=""></deviation></deviation></deviation></category> | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| <category 3=""> <deviation 1=""> <deviation 2=""> <deviation 3=""></deviation></deviation></deviation></category> | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| A subject may have a deviation in more than one category Output: <output name="">, Produced by DATAMAP on ddMnMyyyy hh:mm (CET), SDTM Date: ddMnMyyyy Program: /<folder>/<pre>/<pre>program_name&gt;.sas</pre> <pre>Page x of y</pre></pre></folder></output> | |

Programming notes: Repeat with "Germany", "USA" Show categories as in the PD code list and sort deviations by frequency descending order.

## T DEM

ACT-293987 Protocol: AC-065A309 Summary of baseline demographic characteristics Analysis Set: Safety Analysis Set

| | 200-1000 ug | Uptravi b.i.d. dose<br>200-1000 ug 1200-1600 ug<br>N=xxx N=xxx | |
|---|---|---|---|
| | N=xxx | N=xxx | Total<br>N=xxx |
| Sex [n (%)] | | | |
| Male | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x) |
| Female | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ge [years] | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median<br>Q1, Q3 | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx<br>xx.x<br>xx.xx<br>xx.x<br>xx.x, xx.x | XX, XX |
| ge (years) category [n (%)] | | | |
| < 18 | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x) |
| 18 - 64 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| >= 65 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| eight [cm] | | | |
| n | XX | XX<br>XXX.X<br>XXX.XX<br>XXX.X<br>XXX.X<br>XXX.X | XX |
| Mean | XXX.X | XXX.X | XXX.X |
| SD | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.X | XXX.X | XXX.X |
| Q1, Q3 | xxx.x, xxx.x | xxx.x, xxx.x | XXX.X, XXX. |
| Min, Max | xxx, xxx | xxx, xxx | xxx, xxx |
| ody weight [kg] | | | |
| n<br>Mean | XX | XX<br>VVV V | XX<br>VVV V |
| SD | ^^^. | ^^^ | ^^^. |
| Median | XXX.X | XXX X | XXX.X |
| Q1, Q3 | XXX.X, XXX.X | XXX.X, XXX.X | XXX.X, XXX. |
| Min, Max | xxx, xxx | XX<br>XXX.X<br>XXX.XX<br>XXX.X<br>XXX.X<br>XXX.X | xxx, xxx |
| 4I [kg/m^2] | | | |
| n i | xx | xx | XX |
| Mean | XX.XX | XX.XX | XX.XX |
| SD | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX | XX.XX |
| Q1, Q3 | xx.xx, xx.xx | xx.xx, xx.xx | XX.XX, XX.X |
| Min, Max | XX.X, XX.X | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX, XX.XX | xx.x, xx.x |
| ace [n (%)] | | ( | |
| <race 1=""> <race 2=""></race></race> | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| <race 2=""> <race 3=""></race></race> | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| <race 3=""></race> | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Missing | XXX (XX.X) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x) |
| thnicity [n (%)] | | | |
| <ethnicity 1=""></ethnicity> | xxx (xx.x) | xxx (xx.x) | xxx (xx x) |
| <ethnicity 2=""></ethnicity> | | XXX (XX.X) | XXX (XX X) |
| Missing | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| ountry [n (%)] | | | |
| <country 1=""></country> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| <country 2=""></country> | | | |

SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Programming note: Show race, ethnicity and Countries in descending order of frequency. Show 'Missing' category only if it occurred.


Statistical Analysis Plan Doc No D-18.239

## T AGECATEU

ACT-293987 Protocol: AC-065A309 EudraCT age categories Analysis Set: Safety Analysis Set

| | Uptravi b.i.d. dose | | |
|---|---|---|---|
| | 200-1000 ug<br>N=xxx | 1200-1600 ug<br>N=xxx | Total<br>N=xxx |
| Age (years) category [n (%)] | | | |
| 18 - 64 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 65 - 84 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| >= 85 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
# T BAS

ACT-293987 Protocol: AC-065A309 Summary of baseline disease characteristics Analysis Set: Safety Analysis Set

| | Uptravi b | | |
|---|---|---|---|
| | | 200-1000 ug 1200-1600 ug | |
| | N=xxx | N=xxx | N=xxx |
| Time since diagnosis of PAH [months] | | | |
| n | xx | xx | XX |
| Mean | xx.x | xx.x | XX.X |
| SD | xx.xx | xx.xx | XX.XX |
| Median | xx.x | xx.x | XX.X |
| 01, 03 | XX.X, XX.X | xx.x, xx.x | XX.X, XX. |
| Min, Max | xx, xx | xx, xx | xx, xx |
| AH etiology [n (%)] | | | |
| Idiopathic PAH | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| Heritable PAH | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| Drug or toxin induced PAH | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| PAH associated with | | (, | ( |
| Connective tissue disease | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| HIV infection | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| Portal hypertension | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| Congenital heart disease | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| Schistosomiasis | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| otravi dose at screening [ug b.i.d.] | | | |
| 200 | xxx (xx.x) | | xxx (xx. |
| 400 | xxx (xx.x) | | xxx (xx. |
| 600 | xxx (xx.x) | | xxx (xx. |
| 800 | xxx (xx.x) | | xxx (xx. |
| 1000 | xxx (xx.x) | | xxx (xx. |
| 1200 | , , | xxx (xx.x) | xxx (xx. |
| 1400 | | xxx (xx.x) | xxx (xx. |
| 1600 | | xxx (xx.x) | xxx (xx. |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| HO functional class [n (%)] | | | |
| I | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| II | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx. |
| III | 1 1 | xxx (xx.x) | xxx (xx. |
| III | xxx (xx.x) | XXX (XX.X) | |

Program: /<folder>/program\_name>.sas
Page x of y

Programming note: Show all CRF categories, even if empty. Show 'Missing' category only if it occurred.

## T MH SOC

ACT-293987 Protocol: AC-065A309 <Table Title> Analysis Set: Safety Analysis Set

| System Organ Class | | .i.d. dose | |
|---|---|---|---|
| Preferred Term | 200-1000 ug<br>N=xxx | 1200-1600 ug<br>N=xxx | Total<br>N=xxx |
| Subjects with at least one <pre><pre>cous</pre> disease or</pre> | | | |
| diagnosis | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <system 1="" class="" organ=""></system> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 1="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 3="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 4="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <pre><system 2="" class="" organ=""></system></pre> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <pre><preferred 1="" term=""></preferred></pre> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 3="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 4="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | |
| System Organ Classes and Preferred Terms are base | | | |
| Output: <output name="">, Produced by DATAMAP on ddl</output> | MMyyyy hh:mm (CET) | , | |

SDTM Date: ddMMyyyyy Program: /<folder>/program\_name>.sas Page x of y

Programming note: Sort by descending frequency in the SOC and then by descending frequency and then alphabetically in the PTs. Adapt first line in shell (previous/study concomitant).

#### T CM

ACT-293987 Protocol: AC-065A309 <Table Title> Analysis Set: Safety Analysis Set Period 1: Uptravi, pre-treatment period

| ATC Class | Uptravi b | .i.d. dose | |
|---|---|---|---|
| Preferred Term | 200-1000 ug | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| Subjects with at least one <ongoing> therapy</ongoing> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <atc 1="" class=""></atc> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 1="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 3="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 4="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <atc 2="" class=""> <preferred 1="" term=""> <preferred 2="" term=""> <preferred 3="" term=""> <preferred 4="" term=""></preferred></preferred></preferred></preferred></atc> | XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X) | XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X) | XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X)<br>XXX (XX.X) |
| Preferred Terms are based on WHO-DRUG dictionary The summary does not include PAH-specific therap Output: <output name="">, Produced by DATAMAP on do SDTM Date: ddMMyyyy Program: /<folder>/<pre>/<pre>/<pre>program.onme&gt;.sas Page x of y</pre></pre></pre></folder></output> | oies. | | |

Programming note: Sort by descending frequency in the ATC class in total and then by descending frequency and then alphabetically in the PTs. Display Period line only where applicable. Use the following labels for the concomitant medication table:

| Analysis<br>Period | Label in summary table |
|---|---|
| Screening | Screening Period |
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 1&2 | Period 1 & 2: Uptravi, pre-treatment period and i.v. selexipag treatment period combined |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |
| 1&2&3&FU | Period 1 & 2 & 3: All post-baseline periods including safety follow-up period |

Programming note: Use ATC level 4 for ATC class. Sort by descending frequency in the ATC class and then by descending frequency and then alphabetically in the PTs. Modify first line according to table (previous, ongoing, ...).

#### $T_{CMPAH}$

ACT-293987 Protocol: AC-065A309 Summary of ongoing PAH specific therapies at baseline Analysis Set: Safety Analysis Set

| Number of PAH specific therapies | Uptravi k | o.i.d. dose | |
|---|---|---|---|
| PAH medication category Preferred term | 200-1000 ug<br>N=xxx | 1200-1600 ug<br>N=xxx | Total<br>N=xxx |
| Subjects taking Uptravi | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects with at least one additional PAH specific therapy on top of Uptravi ERA <preferred 1="" term=""> <preferred 2="" term=""> PDE5-Inhibitors <preferred 1="" term=""> <preferred 2="" term=""></preferred></preferred></preferred></preferred> | XXX (XX.X)<br>XXX (XX.X) | XXX (XX.X)<br>XXX (XX.X) | XXX (XX.X)<br>XXX (XX.X) |
| ERA + PDE5 Inhibitors <preferred 1="" term=""> + <preferred 2="" term=""></preferred></preferred> | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| <pre><preferred 1="" term=""> + <preferred 3="" term=""></preferred></preferred></pre> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Preferred Terms are based on WHO-DRUG dictionary veroutput: <pre>Output: <output name="">, Produced by DATAMAP on ddMMMySDTM Date: ddMMMyyyy Program: /<folder>/<pre>/<pre>program_name&gt;.sas Page x of y</pre></pre></folder></output></pre> | | | |

Programming note: Use medication categories based on the PAH specific medication search terms. Sort preferred terms by descending order of frequency. Only show categories which are actually occurring. Continue for triplicate therapies, if occurring.

# $T_EXP_IV$

ACT-293987 Protocol: AC-065A309 Exposure to i.v. selexipag Analysis Set: i.v. Safety Analysis Set

| | Uptravi b. | i.d. dose | |
|---|---|---|---|
| | | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| 37 1 6 1 6 1 1 1 1 (0) 1 | | | |
| Number of infusions received [n (%)] | () | /\ | / |
| 1<br>2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 3 | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| 3 | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) |
| First infusion | | | |
| Planned dose level [uq] | | | |
| 225 (~ 200 p.o.) | xxx (xx.x) | | xxx (xx.x) |
| 450 (~ 400 p.o.) | xxx (xx.x) | | xxx (xx.x) |
| 675 (~ 600 p.o.) | xxx (xx.x) | | xxx (xx.x) |
| 900 (~ 800 p.o.) | xxx (xx.x) | | xxx (xx.x) |
| 1125 (~1000 p.o.) | xxx (xx.x) | | xxx (xx.x) |
| 1350 (~1200 p.o.) | | xxx (xx.x) | xxx (xx.x) |
| 1575 (~1400 p.o.) | | xxx (xx.x) | xxx (xx.x) |
| 1800 (~1600 p.o.) | | xxx (xx.x) | xxx (xx.x) |
| Planned dose [uq] | | | |
| n | XX | XX | XX |
| Mean | xxxx.x | xxxx.x | xxxx.x |
| SD | xxxx.xx | XXXX.XX | XXXX.XX |
| Median | xxxx.x | xxxx.x | xxxx.x |
| Q1, Q3 | xxxx.x, xxxx.x | | xxxx.x, xxxx.x |
| Min, Max | | xxxx, xxxx | xxxx, xxxx |
| Actual dose infused [ug] | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X |
| SD | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXX.X | XXXX.X |
| Q1, Q3 | | XXXX.X, XXXX.X | |
| Min, Max | | xxxx, xxxx | |
| Actual total time of infusion [minutes] | | | |
| n | xx | xx | XX |
| Mean | xx.x | xx.x | xx.x |
| SD | x.xx | x.xx | x.xx |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Second infusion | | | |
| ••• | | | |
| Third infusion | | | |
| SD = Standard deviation Output: <output name="">, Produced by DATAMAP of SDIM Date: ddMMyyyy Program: /<folder>/<pre>/<pre>program_name&gt;.sas Page x of y</pre></pre></folder></output> | n ddMMMyyyy hh:mm | (CET), | |

Programming note: Show all dose categories even if empty, except the 'Other' category which should only be presented if populated.

# $T_EXP_PO$

ACT-293987 Protocol: AC-065A309 Exposure to Uptravi prior to and after i.v. selexipag Analysis Set: <Analysis Set>

| | Uptravi b. | | |
|---|---|---|---|
| | 200-1000 ug<br>N=xxx | 1200-1600<br>ug<br>N=xxx | Total<br>N=xxx |
| Uptravi evening dose before Day 1 [uq] | | | |
| 200 | xxx (xx.x) | | xxx (xx.x) |
| 400 | xxx (xx.x) | | xxx (xx.x) |
| 600 | XXX (XX.X) | | xxx (xx.x) |
| 800<br>1000 | xxx (xx.x)<br>xxx (xx.x) | | xxx (xx.x)<br>xxx (xx.x) |
| 1200 | AAA (AA.A) | xxx (xx.x) | xxx (xx.x) |
| 1400 | | xxx (xx.x) | xxx (xx.x) |
| 1600 | | xxx (xx.x) | xxx (xx.x) |
| Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not received / missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Uptravi morning dose at Day 1 [ug] | , | | , , |
| 200<br>400 | xxx (xx.x) | | xxx (xx.x) |
| 600 | xxx (xx.x)<br>xxx (xx.x) | | xxx (xx.x)<br>xxx (xx.x) |
| 800 | XXX (XX.X) | | xxx (xx.x) |
| 1000 | xxx (xx.x) | | xxx (xx.x) |
| 1200 | | xxx (xx.x) | xxx (xx.x) |
| 1400 | | xxx (xx.x) | xxx (xx.x) |
| 1600<br>Other | () | xxx (xx.x) | xxx (xx.x) |
| Not received / missing | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| - | () | (, | |
| Uptravi evening dose at Day 1 [ug] | 1777 (1777 17) | | 171717 (1717 17) |
| 400 | xxx (xx.x)<br>xxx (xx.x) | | xxx (xx.x)<br>xxx (xx.x) |
| 600 | XXX (XX.X) | | xxx (xx.x) |
| 800 | xxx (xx.x) | | xxx (xx.x) |
| 1000 | xxx (xx.x) | | xxx (xx.x) |
| 1200 | | xxx (xx.x) | xxx (xx.x) |
| 1400<br>1600 | | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| Other | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | XXX (XX.X) |
| Not received / missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Uptravi evening dose at Day 3 [ug] | | | |
| 200 | xxx (xx.x) | | xxx (xx.x) |
| 400 | xxx (xx.x) | | xxx (xx.x) |
| 600 | xxx (xx.x) | | xxx (xx.x) |
| 800 | xxx (xx.x) | | xxx (xx.x) |
| 1000<br>1200 | xxx (xx.x) | 000 (00 o) | XXX (XX.X) |
| 1400 | | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| 1600 | | xxx (xx.x) | xxx (xx.x) |
| Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not received / missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Output: <output name="">, Produced by DATAMAP on d<br/>SDTM Date: ddMMyyyy<br/>Program: /<folder>/<pre>/<pre>program_name&gt;.sas<br/>Page x of y</pre></pre></folder></output> | dMMMyyyy hh:mm (CET), | | |

Programming note: Show all categories even if empty. The 'Other' and 'Not received/missing' categories shall only be shown if populated.

Doc No D-18.239

T\_COMPL\_IV

ACT-293987

Protocol: AC-065A309

Compliance to i.v. selexipag treatment
Analysis Set: i.v. Safety Analysis Set

| | Uptravi b | .i.d. dose | |
|---|---|---|---|
| | 200-1000 ug | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| First infusion | | | |
| FILSC INTUSTON | | | |
| Compliance [%] | | | |
| n | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X |
| SD | xxxx.xx | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXX.X | XXXX.X |
| Q1, Q3 | xxxx.x, xxxx.x | xxxx.x, xxxx.x | xxxx.x, xxxx.x |
| Min, Max | xxxx, xxxx | xxxx, xxxx | xxxx, xxxx |
| Second infusion | | | |
| Compliance [%] | | | |
| n | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X |
| SD | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXX.X | XXXX.X |
| Q1, Q3 | xxxx.x, xxxx.x | xxxx.x, xxxx.x | xxxx.x, xxxx.x |
| Min, Max | xxxx, xxxx | xxxx, xxxx | XXXX, XXXX |
| Third infusion | | | |
| Compliance [%] | | | |
| n | XX | XX | XX |
| Mean | xxxx.x | xxxx.x | xxxx.x |
| SD | xxxx.xx | xxxx.xx | xxxx.xx |
| Median | xxxx.x | xxxx.x | xxxx.x |
| Q1, Q3 | xxxx.x, xxxx.x | xxxx.x, xxxx.x | xxxx.x, xxxx.x |
| Min, Max | xxxx, xxxx | xxxx, xxxx | xxxx, xxxx |
| Overall | | | |
| Compliance [%] | | | |
| n | XX | XX | XX |
| Mean | XXXX.X | XXXX.X | XXXX.X |
| SD | XXXX.XX | XXXX.XX | XXXX.XX |
| Median | XXXX.X | XXXX.X | XXXX.X |
| Q1, Q3 | xxxx.x, xxxx.x | xxxx.x, xxxx.x | xxxx.x, xxxx.x |
| Min, Max | xxxx, xxxx | xxxx, xxxx | XXXX, XXXX |
| Subject with missing infusior<br>SD = Standard deviation<br>Output: <output name="">, Produc<br/>SDTM Date: ddMMMyyyy<br/>Program: /<folder>/<pre>program_r</pre></folder></output> | ced by DATAMAP on ddMMMy | yyy hh:mm (CET), | |

 $\begin{array}{l} T\_EXP\_ADJ \\ \text{ACT-293987} \\ \text{Protocol: AC-065A309} \\ \text{Summary of study treatment administration, reasons for interruptions and end of infusion Analysis Set: i.v. Safety Analysis Set} \end{array}$ 

| • | Uptravi b | .i.d. dose | |
|---|---|---|---|
| | 200-1000 ug | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| First infusion | | | |
| Not received [n (%)] | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Temporary interruptions [n (%)] Due to an AE Not due to an AE | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| End of infusion [n (%)] Premature discontinuation Completed as per protocol | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| Second infusion | | | |
| Not received [n (%)] | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Temporary interruptions [n (%)] Due to an AE Not due to an AE | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| End of infusion [n (%)] Premature discontinuation Completed as per protocol | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| Third infusion | | | |
| Not received [n (%)] | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Temporary interruptions [n (%)] Due to an AE Not due to an AE | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |
| End of infusion [n (%)] Premature discontinuation Completed as per protocol | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |

Subjects may have more than one interruption but are counted only once in each category. Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>//program: /<folder>//program\_name>.sas


#### T PWDT

ACT-293987
Protocol: AC-065A309
Reasons for premature discontinuation of i.v. selexipag treatment Analysis Set: i.v. Safety Analysis Set

| | Uptravi b.: | i.d. dose<br>1200-1600 | |
|---|---|---|---|
| | 200-1000 ug<br>N=xxx<br>n (%) | ug<br>N=xxx<br>n (%) | Total<br>N=xxx<br>n (%) |
| Subjects completed i.v. selexipag treatment | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects prematurely discontinued i.v. selexipag | | | |
| treatment | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | |
| Lost to follow-up | xxx (xx.x) | xxx (xx.x) | |
| Pre-specified discontinuation criteria | xxx (xx.x) | xxx (xx.x) | |
| Subject decision | xxx (xx.x) | xxx (xx.x) | |
| <reason 1=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Physician decision | xxx (xx.x) | xxx (xx.x) | |
| <reason 1=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Sponsor decision | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 1=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <reason 2=""></reason> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>//program\_name>.sas
Page x of y

Programming note: Show all categories written out in the shell in the given order, even if they have zero subjects. Show reason categories as they occurred in descending frequency.

Statistical Analysis Plan Doc No D-18.239

T\_AE\_SOC ACT-293987 Protocol: AC-065A309 <Table title> Analysis Set: <Analysis set>

Period 1: Uptravi, pre-treatment period

| | | | .i.d. dose | | | |
|---|---|---|---|---|---|---|
| | 200-10 | | 1200-1 | | | tal |
| System Organ Class | N=x: | | N=2 | | | XXX |
| Preferred Term | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI |
| Subjects with at least one AE xx | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| <pre><system 1="" class="" organ=""> xx</system></pre> | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| <pre><preferred 1="" term=""> xxx</preferred></pre> | x (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <preferred 2="" term=""> xxx</preferred> | (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X |
| <preferred 3="" term=""> xxx</preferred> | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <preferred 4="" term=""> xxx</preferred> | (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X |
| (System organ class 2> xx: | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| <pre><preferred 1="" term=""> xxx</preferred></pre> | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <preferred 2="" term=""> xxx</preferred> | (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X |
| <preferred 3="" term=""> xxx</preferred> | (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <preferred 4="" term=""> xxx</preferred> | (xx.x) | XX.X, XX.X | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| | | | 1 1 | | | : : |

CI = Confidence interval System Organ Classes and Preferred Terms are based on MedDRA version <xx.x>.

Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),

SDTM Date: ddMMyyyy

Program: /<folder>/program\_name>.sas
Page x of y

Programming note: Sort by descending frequency in the SOC in total and then by descending frequency and then alphabetically in the PTs. Use the following labels:

| Analysis<br>Period | Label in summary table |
|---|---|
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 1&2 | Period 1 & 2: Uptravi, pre-treatment period and i.v. selexipag treatment period combined |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |
| 1&2&3&FU | Period 1 & 2 & 3: All post-baseline periods including safety follow-up period |


Statistical Analysis Plan Doc No D-18.239

T\_AE\_SOC2 ACT-293987 Protocol: AC-065A309 <Table title> Analysis Set: <Analysis set>

| | 200-1000 | _ | 1200-160 | | Total | |
|---|---|---|---|---|---|---|
| | N=xxx | | N=xxx | | N=xxx | ζ |
| MedDRA System organ class<br>Preferred term | Subjects<br>n (%) | Events<br>n | Subjects<br>n (%) | Events<br>n | Subjects<br>n (%) | Events<br>n |
| Subjects with at least one event | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <system 1="" class="" organ=""></system> | xxx (xx.x) | xxx | xxx (xx.x) | xxx | xxx (xx.x) | XXX |
| <preferred 1="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 3="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 4="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <system 2="" class="" organ=""></system> | xxx (xx.x) | xxx | xxx (xx.x) | xxx | xxx (xx.x) | xxx |
| <pre><preferred 1="" term=""></preferred></pre> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 3="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |
| <preferred 4="" term=""></preferred> | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX |

System Organ Classes and Preferred Terms are based on MedDRA version <xx.x>. Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>/program\_name>.sas
Page x of y

Programming note: Table shell for EudraCT/ClinicalTrails.gov disclosure. See Section 7.2.2.1 of the SAP.

T AE PT

ACT-293987 Protocol: AC-065A309 <Table title> Analysis Set: <Analysis set>

Period 1: Uptravi, pre-treatment period

| | 200 1 | Uptravi b | | | | |
|---|---|---|---|---|---|---|
| | | 000 ug - | | .600 ug | | tal |
| | | XXX | | XXX | N= | XXX |
| Preferred term | n (%) | 95% CI | n (%) | 95% CI | n (%) | 95% CI |
| Subjects with at least one AE | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| <pre><preferred 1="" term=""></preferred></pre> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x |
| <pre><preferred 2="" term=""></preferred></pre> | xxx (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X | xxx (xx.x) | XX.X, XX.X |
| <pre><preferred 3="" term=""></preferred></pre> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <pre><preferred 4="" term=""></preferred></pre> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <pre><preferred 5="" term=""></preferred></pre> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| (Preferred term 6> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <pre><preferred 7="" term=""></preferred></pre> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |
| <preferred 8="" term=""></preferred> | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | xx.x, xx.x | xxx (xx.x) | XX.X, XX.X |

CI = Confidence interval
Preferred Terms are based on MedDRA version <xx.x>.
Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),
SDTM Date: ddMMMyyyy
Program: /<folder>/program\_name>.sas
Page x of y

Programming note: Sort by descending frequency and then alphabetically in the PTs in total. Use the following labels:

| Analysis<br>Period | Label in summary table |
|---|---|
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 1&2 | Period 1 & 2: Uptravi, pre-treatment period and i.v. selexipag treatment period combined |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |
| 1&2&3&FU | Period 1 & 2 & 3: All post-baseline periods including safety follow-up period |

Statistical Analysis Plan Doc No D-18.239

# $T\_AE\_PT\_INT$

ACT-293987

Protocol: AC-065A309

Incidence of adverse events by preferred term and maximum intensity Analysis Set: <Analysis set>

| | Uptravi b | | |
|---|---|---|---|
| | 200-1000 ug | 1200-1600 ug | Total |
| Preferred Term | N=xxx | N=xxx | N=xxx |
| Intensity | n (%) | n (%) | n (%) |
| Subjects with at least one AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Mild | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Moderate | XXX (XX.X) | xxx (xx.x) | xxx (xx.x) |
| Severe | XXX (XX.X) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 1="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <preferred 2="" term=""></preferred> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| The maximum intensity of the AE is shown. All post-baseline AEs are shown (Period 1 & 2 & 3 including spreferred Terms are based on MedDRA version <xx.x>. Output: <output name="">, Produced by DATAMAP on ddMMyyyy hh:mmsDTM Date: ddMMyyyyy Program: /<folder>/<pre>/<pre>/<pre>program_name&gt;.sas Page x of y</pre></pre></pre></folder></output></xx.x> | | | |

Programming note: Sort by descending frequency and then alphabetically in the PTs. Show missing category only if it occurred in the data.

# $T\_AEINJ$

ACT-293987

Protocol: AC-065A309

Grade and diagnosis criteria of injection site reactions

Analysis Set: i.v. Safety Analysis Set

| | | b.i.d. dose | |
|---|---|---|---|
| | 200-1000 ug | | Total |
| | N=xxx | N=xxx | N=xxx |
| | n (%) | n (%) | n (%) |
| Subjects with at least one injection site reaction | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects with at least one clinically significant injection site reaction | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Worst Grade<br>Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | | xxx (xx.x) |
| Potentially life threatening | XXX (XX.X) | | |
| rocentrally file enreacening | 71711 (7171-71) | 2222 (222.22) | 71771 (7171-71) |
| Criteria | | | |
| Pain | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Tenderness | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Erythema/redness | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Swelling | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Induration | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Injection site hemorrhage | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

A subject may have more than one diagnosis criterion.

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/<program\_name>.sas

Page x of y

Programming note: For each subject, display the worst grade of all injection site reactions. Display each subject once for all diagnosis criteria reported in a subject.


Statistical Analysis Plan Doc No D-18.239

#### T LB SUM

ACT-293987 Protocol: AC-065A309 <Table Title>

Analysis Set: Safety Analysis Set

Parameter: Haemoglobin [g/L]

| Treatment group | | | Base | eline | | | | Tir | ne Point | | | | Change : | from basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point | n | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max |
| Uptravi b.i.d. dose | 200_1 | 000 110 (1 | .T—xxxxx \ | | | | | | | | | | | | | |
| Baseline | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| Visit 2 Day 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Uptravi b.i.d. dose | 1200- | 1600 ug | (N=xxx) | | | | | | | | | | | | | |
| Baseline | XX | xxx.x | XX.XX | xxx.x | XXX | XXX | | | | | | | | | | |
| Visit 2 Day 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Total (N=xxx) | | | | | | | | | | | | | | | | |
| Baseline | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| Visit 2 Day 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 3 | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |

Baseline is the Day 1 assessment or last assessment prior to Day 1.  $SD = Standard\ deviation$  Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),

SDTM Date: ddMMyyyyy
Program: /<folder>//program name>.sas
Page x of y

Programming note: Continue for all Hematology/Clinical chemistry parameters as stated in Section 7.4 of the SAP.

Statistical Analysis Plan Doc No D-18.239

# $T\_LB\_ABN$

ACT-293987

Protocol: AC-065A309

Incidence of marked laboratory values, by period Analysis Set: Safety Analysis Set

Period 2: i.v. selexipag, treatment period

| | | | Uptravi b | .i.d. dose | |
|---|---|---|---|---|---|
| | | | 200-1000 ug | 1200-1600 ug | Total |
| Category | | | N = xxx | N = xxx | N = xxx |
| Parameter | Grade | Severity of abnormality | n / m (%) | n / m (%) | n / m (%) |
| Hematology | | | | | |
| Hemoglobin | LL | < 100 g/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 80 g/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | Increase > 20 g/L above baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | Increase > 40 g/L above baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Hematocrit | LL | < 0.28 L/L [f], < 0.32 L/L [m] | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 0.2 L/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 0.55 L/L [f], > 0.60 L/L [m] | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 0.65 L/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Platelet count | LL | < 75 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 50 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 600 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 999 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Leukocytes | LL | < 3.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 2.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 20.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 100.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Neutrophils | LL | < 1.5 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| - | LLL | < 1.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Eosinophils | НН | > 5.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Lymphocytes | LL | < 0.8 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 0.5 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 4.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |

| Selexipag (ACT 2939 | 87) |
|------------------------|-----|
| Study AC-065A309 | |
| 2 July 2018, page 89/1 | 35 |


| Statistical Analysis Plan |
|---------------------------|
| Doc No D-18.239 |

| | ннн | > 20.0 x10^9/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
|---|---|---|---|---|---|
| Biochemistry | | | | | |
| ALT | HH | > 3 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| AST | НН | > 3 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Alkaline phosphatase | HH | > 2.5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Total bilirubin | HH | > 2 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HHH | > 5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Creatinine | НН | > 1.5 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 3 xULN | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Sodium | LLL | < 130 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 150 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | ННН | > 155 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Potassium | LL | < 3.2 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | LLL | < 3.0 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | > 5.5 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HHH | > 6.0 mmol/L | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |

ULN = Upper limit of normal. Subjects are summarized in each category they fall into. n = Subjects with event, m = Subjects with assessment in the specified time period (at risk)

Post-baseline abnormalities not present at baseline or abnormalities worsening after baseline are shown.

Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET),

SDTM Date: ddMMyyyyy

Program: /<folder>/program\_name>.sas

Page x of y

# Programming note: Use the following labels:

| Analysis<br>Period | Label in summary table |
|---|---|
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |

Statistical Analysis Plan Doc No D-18.239

## T VS SUM

ACT-293987

Protocol: AC-065A309 Summary and change from baseline of vital signs, by visit Analysis Set: Safety Analysis Set

Parameter: Systolic blood pressure [mmHg]

| Treatment group | | | Base | line | | | | Ti | me Point | | | | Change | from basel | Line | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point | n | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max |
| Uptravi b.i.d. dose 200-10 | 00 ua | (N=xxx) | | | | | | | | | | | | | | |
| Baseline | xx | xxx.x | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| Visit 2 Day 2 + 0 h | XX | xxx.x | XX.XX | xxx.x | xxx | xxx | xxx.x | xx.xx | xxx.x | XXX | xxx | xxx.x | XX.XX | xxx.x | xxx | XXX |
| +25 min | XX | XXX.X | XX.XX | xxx.x | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +87 min | XX | XXX.X | XX.XX | xxx.x | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 2 Day 3 + 0 h | xx | XXX.X | XX.XX | xxx.x | xxx | XXX | xxx.x | xx.xx | xxx.x | XXX | xxx | xxx.x | XX.XX | XXX.X | xxx | XXX |
| +25 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | xxx.x | XX.XX | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX |
| +87 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 3 | XX | xxx.x | XX.XX | xxx.x | XXX | XXX | xxx.x | XX.XX | xxx.x | XXX | XXX | xxx.x | XX.XX | xxx.x | XXX | XXX |
| Uptravi b.i.d. dose 1200-1 | 600 ua | (N=xxx) | | | | | | | | | | | | | | |
| Baseline | XX | XXX.X | xx.xx | xxx.x | XXX | XXX | | | | | | | | | | |
| Visit 2 Day 2 + 0 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | xxx.x | XX.XX | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX |
| | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |

Baseline is the Day 1 assessment or last assessment prior to Day 1. SD = Standard deviation Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET), SDTM Date: ddMMyyyy Program: /<folder>//folder>//sasPage x of y

Programming note: Continue for Total. Then repeat for DBP and pulse.

#### T VS PREDS

ACT-293987 Protocol: AC-065A309 Summary of post-dose values and change from pre-dose of vital signs, by visit Analysis Set: Safety Analysis Set

Parameter: Systolic blood pressure [mmHg]

| Treatment group | | | Pre-dose | e (+0 h) | | | | Ti | me Point | | | | Change | from pre- | dose | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point | n | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max |
| Uptravi b.i.d. dose 200-10 | 000 110 | (N=xxx) | | | | | | | | | | | | | | |
| Visit 2 Day 2 + 0 h | XX | XXX.X | xx.xx | XXX.X | XXX | XXX | | | | | | | | | | |
| +25 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | xx.xx | xxx.x | XXX | XXX | xxx.x | XX.XX | xxx.x | XXX | XXX |
| +87 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| 112 11 | 2121 | 212121 • 21 | 2121 • 2121 | 212221 • 21 | 212121 | 212121 | 212121 • 21 | 7121 • 7121 | 71777.71 | 212121 | 212121 | 212121 • 21 | 7121 • 7121 | 212121 • 21 | 212121 | 21212 |
| Visit 2 Day 3 + 0 h | XX | xxx.x | xx.xx | XXX.X | XXX | XXX | | | | | | | | | | |
| +25 min | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX |
| +87 min | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Uptravi b.i.d. dose 1200- | 1600 110 | (N=xxx) | | | | | | | | | | | | | | |
| Visit 2 Day 2 + 0 h | XX | xxx.x | xx.xx | xxx.x | XXX | XXX | | | | | | | | | | |
| +25 min | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX |
| +87 min | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| 728 11 | | | | | | | | | | | | | | | ***** | **** |
| Visit 2 Day 3 + 0 h | XX | xxx.x | xx.xx | xxx.x | XXX | XXX | | | | | | | | | | |
| +25 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | xxx.x | xx.xx | XXX.X | XXX | XXX | xxx.x | xx.xx | XXX.X | XXX | XXX |
| +87 min | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 4 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 6 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| + 8 h | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| +12 h | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |

SD = Standard deviation
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

| Selexipag (ACT 293987) | | Statistical Analysis Plan |
|--------------------------|--------------|---------------------------|
| Study AC-065A309 | Confidential | Doc No D-18.239 |
| 2 July 2018, page 92/135 | | |

Programming note: Continue for Total. Repeat for DBP and pulse. Show only visits where pre-/post-dose assessments were conducted (Visit 2 Day 2 and Visit 2 Day 3).

#### T VS ABN

ACT-293987

Protocol: AC-065A309

Incidence of marked blood pressure abnormalities, by period

Analysis Set: Safety Analysis Set

Period 2: i.v. selexipag treatment period

| | | | Uptravi b | i.d. dose | |
|---|---|---|---|---|---|
| | | | 200-1000 ug | 1200-1600 ug | Total |
| | | | N = xxx | N = xxx | N = xxx |
| Parameter | Grade | | n / m (%) | n / m (%) | n / m (%) |
| Supine SBP [mmHg] | L | SBP < 90 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | | SBP decrease > 40 from baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | H | 140 <= SBP <= 159 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | | SBP increase > 20 from baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | SBP >= 160 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Supine DBP [mmHg] | L | DBP < 50 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | | DBP decrease > 20 from baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | H | 90 <= DBP <= 99 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | | DBP increase > 20 from baseline | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| | HH | DBP >= 100 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |

SBP = Systolic blood pressure, DBP = Diastolic blood pressure

n = Subjects with event, m = Subjects with assessment in the specified time period (at risk)

Post-baseline abnormalities not present at baseline or abnormalities worsening after baseline are shown.

Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/<program name>.sas

Page x of y

## Programming note: Use the following labels:

| Analysis<br>Period | Label in summary table |
|---|---|
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |

#### T EG SUM

ACT-293987

Protocol: AC-065A309

Summary and change from baseline of quantitative ECG parameters, by visit

Analysis Set: Safety Analysis Set

Parameter: ECG Mean heart rate [bpm]

| Treatment group | | | Base | eline | | | | Ti | me Point | | | | Change | from basel | Line | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point | n | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max |
| Uptravi b.i.d. dose 200-100<br>Baseline | 00 ug<br>xx | (N=xxx)<br>xxx.x | xx.xx | xxx.x | xxx | xxx | | | | | | | | | | |
| Visit 2 Day 2 IV-1 pre<br>IV-1 post | XX<br>XX | xxxxx | XX.XX<br>XX.XX | XXX.X<br>XXX.X | XXX | XXX | XXX.X<br>XXX.X | xx.xx<br>xx.xx | xxx.x | XXX | XXX | xxx.x<br>xxx.x | XX.XX<br>XX.XX | xxx.x | XXX | XXX |
| Visit 2 Day 2 IV-2 pre<br>IV-2 post | XX<br>XX | XXX.X | XX.XX<br>XX.XX | XXX.X<br>XXX.X | XXX | XXX | XXX.X<br>XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X<br>XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 2 Day 3 IV-3 pre<br>IV-3 post | XX<br>XX | XXX.X | XX.XX<br>XX.XX | XXX.X<br>XXX.X | XXX | XXX | XXX.X<br>XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X<br>XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 3 | xx | xxx.x | xx.xx | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX | xxx.x | xx.xx | xxx.x | XXX | XXX |
| Uptravi b.i.d. dose 1200-16<br>Baseline | 600 ug<br>xx | (N=xxx) | xx.xx | xxx.x | xxx | xxx | | | | | | | | | | |
| Visit 2 Day 2 IV-1 pre<br>IV-1 post | XX<br>XX | XXX.X | XX.XX<br>XX.XX | XXX.X<br>XXX.X | XXX | XXX | xxx.x<br>xxx.x | xx.xx | XXX.X<br>XXX.X | XXX | XXX | xxx.x<br>xxx.x | xx.xx<br>xx.xx | XXX.X<br>XXX.X | XXX | XXX |
| ••• | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |

Baseline is the Day 1 assessment or last assessment prior to Day 1.

pre = pre-dose assessment prior to infusion, post = post dose assessment (within 30 minutes after end of infusion)

SD = Standard deviation

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/<program\_name>.sas

Page x of y

Programming note: Continue for Total. Then repeat for PR Interval Single Beat [msec]; QRS Duration, Single Beat [msec]; QT Interval, Single Beat [msec]; QTcB Interval, Single Beat [msec]; QTcF Interval, Single Beat [msec].

Statistical Analysis Plan Doc No D-18.239

#### T EG PREDS

ACT-293987

Protocol: AC-065A309

Summary of post-dose values and change from pre-dose of quantitative ECG parameters, by visit

Analysis Set: Safety Analysis Set

Parameter: ECG Mean heart rate [bpm]

| Treatment group | | | Pre- | dose | | | | Ti | me Point | | | | Change | from pre-c | lose | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point | n | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max | Mean | SD | Median | Min | Max |
| Uptravi b.i.d. dose 200-100 | 0 ug | (N=xxx) | | | | | | | | | | | | | | |
| Visit 2 Day 2 IV-1 pre | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| IV-1 post | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 2 Day 2 IV-2 pre | XX | xxx.x | xx.xx | xxx.x | XXX | xxx | | | | | | | | | | |
| IV-2 post | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Visit 2 Day 3 IV-3 pre | XX | xxx.x | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| IV-3 post | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| Uptravi b.i.d. dose 1200-16 | 00 ug | (N=xxx) | | | | | | | | | | | | | | |
| Visit 2 Day 2 IV-1 pre | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | | | | | | | | | | |
| IV-1 post | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX | XXX.X | XX.XX | XXX.X | XXX | XXX |
| ••• | XX | XXX.X | XX.XX | XXX.X | XXX | XXX | xxx.x | XX.XX | XXX.X | XXX | XXX | xxx.x | XX.XX | XXX.X | XXX | xxx |

pre = pre-dose assessment prior to infusion, post = post dose assessment (within 30 minutes after end of infusion) SD = Standard deviation

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy
Program: /<folder>//program\_name>.sas

Page x of y

Programming note: Continue for Total. Then repeat for PR Interval Single Beat [msec]; QRS Duration, Single Beat [msec]; QT Interval, Single Beat [msec]; QTcB Interval, Single Beat [msec]; QTcF Interval, Single Beat [msec].

Statistical Analysis Plan Doc No D-18.239

## T EG ABN

ACT-293987

Protocol: AC-065A309

Incidence of ECG abnormalities - QT prolongation, by period

Analysis Set: Safety Analysis Set

Period 2: i.v. selexipag treatment period

| | Uptravi b | .i.d. dose | |
|---|---|---|---|
| | 200-1000 ug | 1200-1600 ug | Total |
| | N=xxx | N=xxx | N=xxx |
| Parameter | n / m (%) | n / m (%) | n / m (%) |
| QTc (Bazett's correction), [msec] | | | |
| Value > 450 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 480 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 500 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Increase from baseline > 30 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Increase from baseline > 60 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 450 and increase from baseline > 30 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 450 and increase from baseline > 60 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| QTc (Fridericia's correction), [msec] | | | |
| Value > 450 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 480 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 500 # | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Increase from baseline > 30 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Increase from baseline > 60 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value > 450 and increase from baseline > 30 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Value $>$ 450 and increase from baseline $>$ 60 | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |

n = Subjects with event, m = Subjects with QTc evaluation (at risk)

SDTM Date: ddMMMyyyy

Program: /<folder>/<program name>.sas

Page x of y

<sup>#</sup> Baseline value below treshold OR baseline value above treshold and post baseline value worsened (increased)

If more than one ECG in a period has the same abnormality category, the subject is counted only once.

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),


Statistical Analysis Plan Doc No D-18.239

Programming note: Use the following labels:

| Analysis<br>Period | Label in summary table |
|---|---|
| 1 | Period 1: Uptravi, pre-treatment period |
| 2 | Period 2: i.v. selexipag, treatment period |
| 3&FU | Period 3: Uptravi, post-treatment period including safety follow-up period |
| 2&3&FU | Period 2 & 3: i.v. selexipag, treatment period and Uptravi, post-treatment period including safety follow-up period combined |

# $T\_EG\_QUAL$

ACT-293987

Protocol: AC-065A309

Summary of qualitative ECG findings, by visit Analysis Set: Safety Analysis Set

| | Uptravi b | .i.d. dose | |
|---|---|---|---|
| Visit | 200-1000 ug | 1200-1600 ug | Total |
| Interpreation | N=xxx | N=xxx | N=xxx |
| Finding | n / m (%) | n / m (%) | n / m (%) |
| Baseline/Visit 2 Day 1 | | | |
| Normal | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Unable to interpret | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Abnormal | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 1=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 2=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 3=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 4=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Visit 2 Day 2 IV-1 pre | | | |
| Normal | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Unable to interpret | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Abnormal | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 1=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 2=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 3=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| <finding 4=""></finding> | xxx / xxx (xx.x) | xxx / xxx (xx.x) | xxx / xxx (xx.x) |
| Visit 2, Day 2 IV-1 post | | | |
| Any time post baseline | | | |
| Baseline is the Day 1 assessment or last assessment prior to pre = pre-dose assessment prior to infusion, post = post do n = Subjects with event, m = Subjects with qualitative eval Findings not present at baseline are shown at post baseline Output: <output name="">, Produced by DATAMAP on ddMMMyyyy hh:</output> | ase assessment (within 30 minutes amuation (at risk in category) timepoints. | fter end of infusion) | |

Statistical Analysis Plan Doc No D-18.239

Program: /<folder>/program\_name>.sas
Page x of y

Programming note: Continue for all scheduled ECG assessments (Visit 2 Day 2 IV-2 pre/post, Visit 2 Day 3 IV3 pre/post, Visit 3) and for any time post baseline. Sort abnormalities by descending total incidence.

# $T_WHO_SUM$

ACT-293987

Protocol: AC-065A309

Summary of WHO functional class, by visit

Analysis Set: Safety Analysis Set

| | Untravi h | .i.d. dose | |
|---|---|---|---|
| | 200-1000 ug | 1200-1600 ug | Total |
| Visit. | N=xxx | N=xxx | N=xxx |
| WHO functional class | n (%) | n (%) | n (%) |
| wild fullectional class | 11 (0) | 11 (0) | 11 (0) |
| Baseline | | | |
| WHO FC T | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | |
| Visit 2 Day 3 | | | |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| TT: -: + 2 | | | |
| Visit 3<br>WHO FC I | ( | ( | ( |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |
| Missing | XXX (XX.X) | xxx (xx.x) | |
| riissiiig | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) |
| Worst post baseline (including unscheduled visits) | | | |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 3 | , , , | , , | , , |
| Best post baseline (including unscheduled visits) | | | |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Baseline is the Day 1 assessment or last assessment production of the Day 1 assessment production of th | | | |

Programming note: The missing category will only be presented if occurring in the data.

 $T_WHO_CHG$ 

ACT-293987

Protocol: AC-065A309

Shift table of WHO functional class from baseline to each study visit

Analysis Set: Safety Analysis Set

Treatment group: Uptravi b.i.d. dose 200-1000 ug (N=xxx)

| | | | Baseline | | |
|---|---|---|---|---|---|
| Visit<br>WHO functional | WHO FC I | WHO FC II | WHO FC III | WHO FC IV | Missing |
| class | n (%) | n (%) | n (%) | n (%) | n (%) |
| Visit 2 Day 3 | , , | , , | | , , | , , |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Visit 3 | | | | | |
| VISIC 3<br>WHO FC T | / | /\ | / | / | / |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | | xxx (xx.x) | | xxx (xx.x) | xxx (xx.x) |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Worst post-baseline | (including une | cheduled visits) | | | |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IT | xxx (xx.x) | xxx (xx.x) | XXX (XX.X) | XXX (XX.X) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | XXX (XX.X) | xxx (xx.x) | XXX (XX.X) | XXX (XX.X) |
| WHO FC TV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX (XX.X) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MISSING | XXX (XX.X) | xxx (xx.x) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Best post-baseline | (including unsc | heduled visits) | | | |
| WHO FC I | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC II | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC III | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WHO FC IV | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Missing | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | / | (/ | / | | () |

Baseline is the Day 1 assessment or last assessment prior to Day 1. Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET), SDTM Date: ddMMyyyyy

Program: /<folder>/program\_name>.sas

Page x of y

Programming note: The missing category will only be presented if occurring in the data. Repeat for Dose >=1200 ug and total groups.

# $T_PK_CON_SUM$

ACT-293987

Protocol: AC-065A309

treatment

Analysis Set: Pharmacokinetic Analysis Set

Dose group: 200 ug b.i.d. p.o./ 225 ug b.i.d. i.v.

| Treatment | | 7 | Comptolic man | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time | | Arithmetic mean | Geometric mean | | | | | |
| point | n | (95% CI) | (95% CI) | SD | SE | Min | Median | Max |
| Uptravi | | | | | | | | |
| 0 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 1 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 2 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 4 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 6 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 8 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 12 h | XXX | xxx ( $xx.x$ , $xx.x$ ) | xxx ( $xx.x$ , $xx.x$ ) | XXX | XXX | XXX | XXX | XXX |
| i.v. selex | ipaq | | | | | | | |
| 0 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 25 min | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | xxx | XXX |
| 87 min | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 4 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 6 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | XXX | XXX |
| 8 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | xxx | XXX |
| 12 h | XXX | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) | XXX | XXX | XXX | xxx | XXX |

 ${\tt CI} = {\tt Confidence}$  interval,  ${\tt SD} = {\tt Standard}$  deviation,  ${\tt SE} = {\tt Standard}$  error, p.o. = per os, b.i.d. = twice daily; i.v. = intravenous

Implausible plasma concentrations are not included in the summary.

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/<program\_name>.sas

Page  ${\tt x}$  of  ${\tt y}$ 

Programming note: Continue for dose groups 400p.o./450i.v., 600p.o./675i.v., 800p.o./900i.v., 1000p.o./1125i.v., 1200p.o./1350i.v., 1400p.o./1575i.v., 1600p.o./1800i.v., and dose normalized.

# $T_PK\_EP\_SUM$

ACT-293987

Protocol: AC-065A309

Summary of PK parameters of <selexipag/ACT-333679> by dose level and treatment Analysis Set: Pharmacokinetic Analysis Set

Dose level: 200 ug b.i.d. p.o./ 225 ug b.i.d. i.v.

| PK parameter<br>Statistic | Uptravi<br>N=xxx | i.v. selexipag<br>N=xxx |
|---|---|---|
| Subjects in dose level | xxx | xxx |
| AUCtau,ss [ng.h/mL] | | |
| N | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| Geometric mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| SD | XX.X | XX.X |
| SE | XXX | XXX |
| CV%<br>CV ln% | XX.X | XX.X |
| Median | xx.x<br>xx.x | xx.x<br>xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Ctrough,ss, Oh [ng/mL] | | |
| n | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| Geometric mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| SD | XX.X | XX.X |
| SE | XXX | XXX |
| CV% | XX.X | XX.X |
| CV ln%<br>Median | XX.X | XX.X |
| Min, Max | xx.x<br>xx.x, xx.x | xx.x<br>xx.x, xx.x |
| Ctrough,ss, 12h [ng/mL] | | |
| n | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| Geometric mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| SD | xx.x | xx.x |
| SE | XXX | XXX |
| CV% | XX.X | XX.X |
| CV ln% | XX.X | XX.X |
| Median | XX.X | XX.X |
| Min, Max | xx.x, xx.x | XX.X, XX.X |
| Cmax,ss [ng/mL]<br>n | xxx | 7777 |
| Arithmetic mean (95% CI) | xxx (xx.x, xx.x) | xxx<br>xxx (xx.x, xx.x) |
| Geometric mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| SD | XXX (XX.X, XX.X)<br>XX.X | XXX (XX.X, XX.X)<br>XX.X |
| SE | XX.X<br>XXX | XXX |
| CV% | XX.X | XX.X |
| CV ln% | XX.X | xx.x |
| Median | XX.X | XX.X |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| tmax,ss [h] | | |
| n | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| SD | XX.X | xx.x |
| SE<br>CV w% | XXX<br>XX.X | xxx<br>xx.x |
| | XX•X | **** |
| Median | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

CI = Confidence interval, SD = Standard deviation, SE = Standard error, CV% = Coefficient of variation [%], CV b% = Between-subject coefficient of variation [%], CV ln% = Coefficient of variation of logarithmized values [%], p.o. = per os, b.i.d. = twice daily, i.v. = intravenous Values obtained from implausible plasma concentrations are not included in the summary. Output: <Output name>, Produced by DATAMAP on ddMMMyyyyy hh:mm (CET), SDTM Date: ddMMMyyyy

Program: /<folder>/<program\_name>.sas

Page x of y

Programming note: Continue for dose all dose levels and dose normalized.

## T PK\_RATIO\_SUM

ACT-293987

Protocol: AC-065A309

Summary of PK parameters of ratio ACT-333679/selexipag concentration by dose level and treatment Analysis Set: Pharmacokinetic Analysis Set

Dose level: 200 ug b.i.d. p.o./ 225 ug b.i.d. i.v.

| PK parameter<br>Statistic | Uptravi<br>N=xxx | i.v. selexipag<br>N=xxx |
|---------------------------|--------------------|-------------------------|
| Subjects in dose level | XXX | XXX |
| AUCtau,ss [ng.h/mL] | | |
| N | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.xx, xx.xx) | xxx (xx.xx, xx.xx) |
| Geometric mean (95% CI) | xxx (xx.xx, xx.xx) | xxx (xx.xx, xx.xx) |
| SD | xx.xxx | xx.xxx |
| SE | XX.XXX | XX.XXX |
| CV% | XX.XX | XX.XX |
| CV ln% | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Min, Max | xx.xx, xx.xx | xx.xx, xx.xx |
| Cmax,ss [ng/mL] | | |
| n | XXX | XXX |
| Arithmetic mean (95% CI) | xxx (xx.xx, xx.xx) | xxx (xx.xx, xx.xx) |
| Geometric mean (95% CI) | xxx (xx.xx, xx.xx) | xxx (xx.xx, xx.xx) |
| SD | XX.XXX | XX.XXX |
| SE | XX.XXX | XX.XXX |
| CV% | XX.XX | XX.XX |
| CV ln% | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Min, Max | XX.XX, XX.XX | XX.XX, XX.XX |

CI = Confidence interval, SD = Standard deviation, SE = Standard error, CV% = Coefficient of variation (SD/mean) [%], CV\_ln% = Coefficient of variation of logarithmized values, [%] p.o. = per os, b.i.d. = twice daily; i.v.= intravenous Values obtained from implausible plasma concentrations are not included in the summary.

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/program\_name>.sas

Page x of y

Programming note: Continue for dose all dose levels and dose normalized.

# *T\_PK\_MM*ACT-293987

Protocol: AC-065A309

dose level

Analysis Set: Pharmacokinetic Analysis Set

| Endpoint<br>Statistic | Cmax,ss | AUCtau ss |
|---|---|---|
| Dose level: 200 ug b.i.d. p.o./ 225 ug | b.i.d. i.v. | |
| n | xxx | XXX |
| Ratio of geom. means (i.v./p.o) | x.xx ( $x.xx$ , $x.xx$ ) | x.xx ( $x.xx$ , $x.xx$ ) |
| 90% CI | x.xxx, x.xxx | x.xxx, x.xxx |
| CV b[%] | xx.xx | XX.XX |
| Dose level: 400 ug b.i.d. p.o./ 450 ug | b.i.d. i.v. | |
| n | XXX | xxx |
| Ratio of geom. means (i.v./p.o) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| 90% CI | x.xxx, x.xxx | xxx (xx.x, xx.x) |
| CV b[%] | xx.x | xx.x |
| Dose level: | | |
| n | xxx | xxx |
| Ratio of geom. means (i.v./p.o) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| 90% CI | x.xxx, x.xxx | xxx (xx.x, xx.x) |
| CV b[%] | XX.X | XX.X |
| Dose level: Normalized dose (200 ug) | | |
| n | XXX | xxx |
| Ratio of geom. means (i.v./p.o) | xxx (xx.x, xx.x) | xxx (xx.x, xx.x) |
| 90% CI | x.xxx, x.xxx | xxx (xx.x, xx.x) |
| CV b[%] | xx.x | XX.X |
| CI = Confidence interval, n.e. = not exintravenous Geometric mean ratios were obtained by of a mixed model with treatment as fix data. CV_b[%] was computed using the m Values obtained from implausible plasm Output: <output name="">, Produced by DAT SDTM Date: ddMMyyyy Program: /<folder>/<pre>/<pre>program_name&gt;.sas</pre></pre></folder></output> | r computing the anti-log of t<br>ted and subject as random eff<br>mean squared error or residua<br>na concentrations are not inc | the treatment group difference fect to the log-transformed als as a measure of variation. |

Programming note: Display all dose levels. For dose levels not sufficiently populated to allow an estimation populate only 'n' row and show 'n.e.' for the remaining statistics.

#### T PK POW

ACT-293987

Protocol: AC-065A309

Dose proportionality of AUCtau of <selexipag/ACT-333679> after i.v. selexipag: Power model

estimation

Analysis Set: Pharmacokinetic Analysis Set

| n | beta | SE (beta) | 90% CI |
|-----|-------|-----------|--------------|
| | | | _ |
| XXX | X.XXX | XX.XXX | x.xxx, x.xxx |

CI = Confidence interval

Dose proportionality will be assumed if beta is close to 1, i.e., if the CI of beta includes 1. Values obtained from implausible plasma concentrations are not included in the analysis.

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/program\_name>.sas

Page x of y

Programming note: Produce table only if sufficient subjects are included in at least three dose levels.


Statistical Analysis Plan Doc No D-18.239

# *T\_PK\_WIL*ACT-293987

Protocol: AC-065A309

Location shift analysis of tmax, ss of <selexipag/ACT-333679>

Analysis Set: Pharmacokinetic Analysis Set

| i.v. selexipag - Uptravi | | | |
|--------------------------|--------|--------------|---------|
| n | Median | 90% CI | p-value |
| xxx | x.xxx | x.xxx, x.xxx | x.xxxx |

CI = Confidence interval from a Hodges - Lehmann estimation. p-value is derived from a Wilcoxon signed rank test.

Values obtained from implausible plasma concentrations are not included in the analysis. Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>/program\_name>.sas Page x of y

F EXP

ACT-293987

Protocol: AC-065A309

Shift in selexipag dose between oral and i.v. treatment

Analysis Set: i.v. Safety Analysis Set



Output: <Output name>, Produced by DATAMAP on ddMMMyyyyy hh:mm (CET),

SDTM Date: ddMMMyyyy

Program: /<folder>/program\_name>.sas

age x of y

Programming note: This is just a conceptual graphic showing subjects from two dose levels (there will be more levels in the study). Adapt to Actelion standards. Jitter series plots such that individual subject lines are clearly visible. Do use color for each series plot.
### F PK POW

ACT-293987

Protocol: AC-065A309

Dose proportionality of AUCtau <selexipag/ACT-333679> after i.v. selexipag: Power model estimation Analysis Set: Pharmacokinetic Analysis Set



Values obtained from implausible plasma concentrations are not included in the analysis. Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program\_ name>.sas

Page x of y

Programming note: This is just a general sketch: Display log dose vs. log AUC and display a regression line from the model with the slope of estimated beta. Add a second line with beta (i.e., slope) =1 as reference.

Statistical Analysis Plan Doc No D-18.239

### L SCRF

ACT-293987
Protocol: AC-065A309
Listing of screening failures
Analysis Set: Screened Analysis Set
Country: <country>, Site: <Site number>

| Subject<br>number | Date | Reason for screening failure |
|---|---|---|
| 1001001<br>1001002 | ddMMyyyy<br>ddMMyyyy | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>//program\_name>.sas
Page x of y

Programming note: Add specification for reason of screening failure, if available from the database.

Statistical Analysis Plan Doc No D-18.239

# L PWDS

ACT-293987 Protocol: AC-065A309 Listing of reasons for premature discontinuation from the study Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Status | Date / Day | Reason for discontinuation from the study | Details |
|---|---|---|---|---|
| 1001001<br>1001002<br>1001003 | Completed Discontinued Discontinued | ddMMyyy / xxx<br>ddMMyyy / xxx<br>ddMMyyy / xxx | Death<br>Physician decision | xxxx xxxxxxxx |

### L PHYS

ACT-293987 Protocol: AC-065A309 Listing of physical examination results Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Visit | Date / Day | Body system | Result | Specify abnormality | Clin.<br>sign. |
|---|---|---|---|---|---|---|
| 1001001 | Screening | ddMMyyy / xxx | General appearance<br>Head, ears, eyes, nose, throat | Normal<br>Abnormal | XXXXXXXXX | No |
| | Visit 2 - Day 1 | ddMMyyy / xxx | ••• | | | |
| | Visit 3 | ddMMyyy / xxx | | | | |
| SDTM Date: | <folder>/<program_name>.</program_name></folder> | | y hh:mm (CET), | | | |

Programming note: Display 'not done' in the result section if a specific physical examination was databased as such.

Statistical Analysis Plan Doc No D-18.239

# L PWDT

ACT-293987 Protocol: AC-065A309 Listing of reasons for premature discontinuation of i.v. selexipag treatment Analysis Set: i.v. Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Status | Reason for discontinuation of i.v. selexipag treatment | Details |
|---|---|---|---|
| 1001001<br>1001002<br>1001003 | Completed<br>Discontinued<br>Discontinued | Death<br>Physician decision | XXXX XXXXXXXX |

L AE

ACT-293987 Protocol: AC-065A309 Listing of <Listing title> Analysis Set: <Analysis set>

Country: <country>, Site: <Site number>

| Subject<br>number | System Organ Class<br>Preferred Term<br>(Reported Term) | Start<br>date/<br>time/Day | End date/<br>time/Day | Duration<br>(days) | Seri<br>ous | Ser.<br>crit. | Inten<br>sity | Concom.<br>trt.<br>given | Action<br>taken i.v.<br>selexipag | Related<br>to i.v.<br>selexipag | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1001001 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMMyyyy/<br>hh:mm/xx | ddMMyyyy/<br>hh:mm/xx | xx | Y | 2,3 | sev | Y | 6 | Y | Revcovered/<br>Resolved |
| 1001002 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMyyyy/<br>hh:mm/xx | ddMMyyyy/<br>hh:mm/xx | xx | N | | mod | N | 6 | N | Revcovering/<br>Resolving |

\$ = Injection site reaction adverse event
Seriousness criteria: 1 Death, 2 Life-threatening, 3 Results in significant disability, 4 Birth defect/congenital anomaly,
5 Required/Prolonged hospitalization, 6 Other medical importance
Action taken with i.v. selexipag: 1 Dose not changed, 2 Dose increased, 3 Dose reduced, 4 Drug interrupted, 5 Drug withdrawn,
6 Not applicable, 7 Unknown
Intensity: mild = Mild, mod = Moderate, sev = Severe
System Organ Classes and Preferred Terms are based on MedDRA version <xx.x>.
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyvyv

SDTM Date: ddMMyyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

# L DTH

ACT-293987 Protocol: AC-065A309 Listing of all deaths Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Death<br>Date / Time / Day | Primary cause of death (Reported term) |
|---|---|---|
| 1001002 | ddMMMyyy / hh:mm / xxx | XXXXXXXX<br>(XXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Preferred Terms are based on MedDRA version <xx.x>.
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

# L AEINJ

ACT-293987 Protocol: AC-065A309 Listing of all injection site reactions Analysis Set: i.v. Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Onset<br>Date / Time / Day | Resolution<br>Date / Time / Day | Criteria | Grade | Clinically<br>Significant | Adverse event<br>Preferred Term |
|---|---|---|---|---|---|---|
| 1001002 | | ddMMMyyy / hh:mm / xxx<br>ddMMMyyy / hh:mm / xxx | Swelling<br>Pain | Moderate<br>Mild | Y<br>N | xxxxxxxx |

Preferred Terms are based on MedDRA version <xx.x>.
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

### L LAB

ACT-293987 Protocol: AC-065A309 Listing of laboratory parameters Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject | Subject St | | | | Reference | Change 1 | Change from baseline |
|---|---|---|---|---|---|---|---|
| number | Parameter [SI Unit] | Visit | Day | Value | Range | Absolute | Percent |
| 1001002 | Hemoglobin [g/L] | Screening | | xxxx | xxx - xxx | XXX | xxx |
| | | Unscheduled | | xxxx H | xxx - xxx | XXX | XXX |
| | | Unscheduled | | xxxx\$ | xxx - xxx | XXX | XXX |
| | | Visit 2 - Dav 1 | | xxxx*HH | xxx - xxx | XXX | XXX |

<sup>\* =</sup> Baseline, H = Above upper limit of normal range, L = Below lower limit of normal range (as flagged by the laboratory)
\$ = Local lab value, not used for summary tables
HH, HHH: Marked abnormally high values, LL, LLL: Marked abnormally low values (derived using SI units)
Newly occurring or worsening post-baseline marked abnormalities are flagged.
Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>/
Program\_name>.sas
Page x of y

 $L_{-}VS$ 

ACT-293987 Protocol: AC-065A309 Listing of vital signs, body weight and height Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Parameter [SI Unit] | Visit | Study<br>Day | Time<br>point | Value | Change from baseline |
|---|---|---|---|---|---|---|
| 1001002 | Systolic blood pressure [mmHg] | Screening<br>Visit 2 - Day 1 | xx<br>xx | Pre dose | xxxx<br>xxxx* | XXXXX |
| | | | | + 25 min<br>+ 87 min<br>+ 4 h | XXXXHH<br>XXXX<br>XXXX | XXXX<br>XXXXX<br>XXXX |

<sup>\* =</sup> Baseline, HH: Marked abnormally high values, LL: Marked abnormally low values Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET), Newly occurring or worsening post-baseline marked abnormalities are flagged. SDTM Date: ddMMyyyy Program: /<folder>/
//folder>/
//folder>/
// Sas Page x of y

Selexipag (ACT 293987) **Study AC-065A309** 2 July 2018, page 119/135

### Confidential

Statistical Analysis Plan Doc No D-18.239

# L PD

ACT-293987 Protocol: AC-065A309 Listing of protocol deviations Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Category | Identifier | Description | Exclusion from<br>PKS | Important<br>PD |
|---|---|---|---|---|---|
| 1001002 | Screening period | 000 | XXXXXXXXXXXXXXX | Yes | Yes |
| | Treatment and observation period | 000 | YYYYYYYYYYYYYYY | No | No |

Statistical Analysis Plan Doc No D-18.239

# $L\_ANSET$

ACT-293987 Protocol: AC-065A309 Listing of analysis sets Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Screened<br>analysis set (SCR) | Safety<br>analysis set (SAF) | i.v. Safety<br>analysis set (ivSAF) | Pharmacokinetic<br>analysis set (PKS) | Reason |
|---|---|---|---|---|---|
| 1001001 | Yes | No | No | No | Not treated with i.v. selexipag |
| 1001002 | Yes | Yes | Yes | No | XXXXX |

Statistical Analysis Plan Doc No D-18.239

# L DEM

ACT-293987 Protocol: AC-065A309 Listing of demographics Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Age<br>[years] | Sex | Race | Ethnicity | Weight<br>[kg] | Height<br>[cm] | BMI<br>[kg/m^2] |
|---|---|---|---|---|---|---|---|
| 1001001 | 23 | M | White | Hispanic or Latino | 81.1 | 180 | 25.0 |
| 1001002 | 65 | F | Other: xxxxx | Not Hispanic or Latino | 74.2 | 163 | 27.9 |

Selexipag (ACT 293987) **Study AC-065A309** 2 July 2018, page 122/135

### Confidential

Statistical Analysis Plan Doc No D-18.239

# L BAS

ACT-293987 Protocol: AC-065A309 Listing of baseline disease characteristics Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Date of initial PAH<br>diagnosis | Months since initial diagnosis at baseline | Etiology of PAH | PAH associated with | Uptravi dose at screening [ug bid] | WHO functional class |
|---|---|---|---|---|---|---|
| 1001001 | ddMMyyyy | XX.X | Idiopathic PAH | | 800 | II |
| 1001002 | ddMMyyyy | XX.X | PAH associated with | Connective tissue | 1200 | III |

Statistical Analysis Plan Doc No D-18.239

L MH

ACT-293987 Protocol: AC-065A309 Listing of medical history Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | System Organ Class<br>Preferred Term<br>(Reported Term) | Start date | End date | Ongoing at<br>Screening |
|---|---|---|---|---|
| 1001001 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMyyyy | ddMMyyyy | |
| 1001002 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMyyyy | | Yes |

System Organ Classes and Preferred Terms are based on MedDRA version <xx.x>. Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET), SDTM Date: ddMMyyyy Program: /<folder>/program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

L CM

ACT-293987 Protocol: AC-065A309 <Title>

Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | ATC Class<br>Preferred Term<br>(Reported Term) | Start date /<br>Day | End date /<br>Day | Start<br>in<br>Period | End in<br>Period | Started prior to start of i.v. selexipag? | Ongoing<br>at End<br>of<br>Study | Dose/Unit/Frequency/Indication/Route |
|---|---|---|---|---|---|---|---|---|
| 1001001 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMyyyy/xx | ddMMyyyy/xx | | 1 | Yes | No | 25/mg/bid/XXXXXX/Oral |
| 1001002 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ddMMyyyy/xx | | FU | | No | Yes | XXXX/XXX/XXXX/XXXXXXXXXXXXXXXXXXXXXXXX |

ATC Classes and Preferred Terms are based on WHO-DRUG dictionary version <xxx>.
# PAH specific medication
[1] Previous therapy, [2] Ongoing therapy, [3] Study concomitant therapy
Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

# $L_{EXP\_PO}$

ACT-293987 Protocol: AC-065A309 Listing of Uptravi dosing records Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject number | Time point | Uptravi<br>administered | Date/time | Uptravi dose [ug] |
|---|---|---|---|---|
| 1001001 | Evening before Day 1<br>Day 1 - Morning<br>Day 1 - Evening<br>Day 3 - Evening | No | ddMMyyyy/hh:mm<br>ddMMyyyy/hh:mm<br>ddMMyyyy/hh:mm | 800<br>800<br>600 |

1001002

Statistical Analysis Plan Doc No D-18.239

# $L\_{EXP\_IV}$

ACT-293987 Protocol: AC-065A309 Listing of study treatment dosing records Analysis Set: i.v. Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Time point/<br>Visit | Start date/time | End date/time | Duration<br>[min] | Concentration<br>[ug/mL] | Infusion rate<br>[mL/h] | Reason for change/end |
|---|---|---|---|---|---|---|---|
| 1001001 | Day 2 morning<br>Day 2 evening | ddMMMyyyy/hh:mm<br>ddMMMyyyy/hh:mm | ddMMMyyyy/hh:mm<br>ddMMMyyyy/hh:mm | XX | 22.5<br>22.5 | 20<br>37.5 | Infusion rate change<br>Temporarily interrupted due to<br>an AE |
| | Day 3 morning | ddMMMyyyy/hh:mm | ddMMMyyyy/hh:mm | XX | 22.5 | 20 | Completed as per protocol |

1001002

Statistical Analysis Plan Doc No D-18.239

L COMP

ACT-293987 Protocol: AC-065A309 Listing of compliance with i.v. selexipag treatment Analysis Set: i.v. Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject number | Time point/<br>Visit | Planned dose<br>[ug] | Actual dose [ug] | Compliance [%] |
|---|---|---|---|---|
| 1001001 | Day 2 morning<br>Day 2 evening<br>Day 3 morning<br>Overall | 900<br>900<br>900 | 850<br>870<br>900 | 94.4<br>96.7<br>100.0<br>97.0 |

1001002

### L EG

ACT-293987 Protocol: AC-065A309 Listing of quantitative ECG measurements Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Visit / Time<br>point | Date/time | Heart rate<br>[bpm] | RR<br>[ms] | PR<br>[ms] | QRS<br>[ms] | QT<br>[ms] | QTcB<br>[ms] | QTcF<br>[ms] |
|---|---|---|---|---|---|---|---|---|---|
| 1001002 | Visit 2 - Day 1 | ddMMMyyyy/hh:mm | xx* | xxx* | xxx* | xxx* | xxx* | xxx* | xxx* |
| 1001002 | Unscheduled | ddMMyyyy/hh:mm | XX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Visit 2 - Day 2 IV-1 pre-dose | ddMMyyyy/hh:mm | XX | XXX | XXX | XXX | XXX | XXX | XXX |
| | Visit 2 - Day 2 IV-1 post-dose | ddMMMyyyy/hh:mm | XX | XXX | XXX | xxx | XXX | xxx # | XXX |
| | Visit 2 - Day 2 IV-2 pre-dose | ddMMMyyyy/hh:mm | xx # | XXX | xxx # | XXX | XXX | XXX | XXX |
| | Visit 2 - Day 2 IV-2 post-dose | ddMMMyyyy/hh:mm | XX | XXX | XXX | XXX | XXX | xxx # | XXX |
| | Visit 2 - Day 3 IV-3 pre-dose | ddMMMyyyy/hh:mm | xx | XXX | xxx # | XXX | XXX | XXX | XXX |
| | Visit 2 - Day 3 IV-3 post-dose | ddMMMyyyy/hh:mm | xx | XXX | XXX | XXX | XXX | XXX | XXX |
| | Visit 3 | ddMMMvvvv/hh:mm | xx | XXX | XXX | XXX | XXX | XXX | XXX |

QTcB = QT interval Bazett's correction, QTcF = QT interval Fridericia's correction \* = Baseline, # = Marked abnormal value
Newly occurring or worsening post-baseline marked abnormalities are flagged.
Output: <Output name>, Produced by DATAMAP on ddMMyyyyy hh:mm (CET),
SDTM Date: ddMMyyyyy
Program: /<folder>//Program\_name>.sas
Page x of y

Statistical Analysis Plan Doc No D-18.239

# $L\_EG\_QUAL$

ACT-293987 Protocol: AC-065A309 Listing of qualitative ECG findings Analysis Set: Safety Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Visit / Time<br>point | Date/time | Interpretation | Findings |
|---|---|---|---|---|
| 1001002 | Visit 2 - Day 1 Unscheduled Visit 2 - Day 2 IV-1 pre-dose Visit 2 - Day 2 IV-1 post-dose Visit 2 - Day 2 IV-2 pre-dose Visit 2 - Day 2 IV-2 post-dose Visit 2 - Day 3 IV-3 pre-dose Visit 2 - Day 3 IV-3 post-dose Visit 2 - Day 3 IV-3 post-dose Visit 3 | ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMyyyy/hh:mm ddMMfyyyy/hh:mm ddMMfyyyy/hh:mm ddMMfyyyy/hh:mm | Normal Abnormal Normal Normal Normal Normal Normal Normal Normal | XXXX |

Output: <Output name>, Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy Program: /<folder>//program\_name>.sasPage x of y

Programming note: Layout may change with the structure of the data.

Statistical Analysis Plan Doc No D-18.239

# L WHO

ACT-293987 Protocol: AC-065A309 Listing of WHO functional class Analysis Set: Screened Analysis Set

Country: <country>, Site: <Site number>

| Subject<br>number | Visit | WHO functional class |
|---|---|---|
| 1001003 | Screening<br>Visit 2 - Day 1<br>Visit 2 - Day 3<br>Unscheduled<br>Visit 3 | II<br>II*<br>III<br>I |

The Baseline Output: Output: Output: Coutput name, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMMyyyy
Program: /<folder>//program\_name.sas
Page x of y

# L PK CONC

Page x of y

ACT-293987 Protocol: AC-065A309 Listing of selexipag / ACT-333679 plasma concentrations Analysis Set: Pharmacokinetic Analysis Set

| 1001002 Visit 2 Visit 2 | - | Pre-dose 1 h post-dose 2 h post-dose | XXX #<br>XXX<br>XXX | xxx #<br>xxx<br>xxx |
|---|---|---|---|---|
| Visit 2 | | | | |
| | | Pre-infusion start 5 min post infusion start 7 min post infusion start 4 h post infusion start | XXX #<br>XXX<br>XXX<br>XXX # | xxx #<br>xxx<br>xxx<br>xxx<br>xxx # |

Programming note: List by subject. Only list subjects who provided data. Layout may change slightly depending upon data structure.

### L PK DER

ACT-293987 Protocol: AC-065A309 Listing of derived PK parameters of selexipag and ACT-333679

Analysis Set: Pharmacokinetic Analysis Set

| | | | | i.v. selexip | ag | | Uptravi | | Ratio i.v.<br>Upt | selexipag /<br>cravi |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Subject<br>number | Time point | Dose<br>[ug<br>bid] | Selexipag | ACT-<br>333679 | Dose<br>[ug<br>bid] | Selexipag | ACT-<br>333679 | Selexipag | ACT-333679 |
| Ctrough,ss [ng/mL] | 1001002 | Pre-dose | xxxx | xxx# | xxx# | xxx | xxx | xxx | xxx | xxx |
| | 1001004 | 12 h post-dose<br>Pre-dose<br>12 h post-dose | XXXX<br>XXXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | xxx<br>xxx |
| Dose normalized<br>Ctrough,ss,norm<br>[ng/mL] | 1001002 | Pre-dose | xxxx | XXX | XXX | xxx | XXX | XXX | XXX | xxx |
| [119/1111] | | 12 h post-dose | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Cmax,ss [ng/mL] | 1001002 | | xxxx | xxx | xxx | xxx | XXX | xxx | XXX | XXX |
| Dose normalized Cmax,ss,norm [ng/mL] | 1001002 | | | XXX | XXX | | xxx | xxx | xxx | XXX |
| AUCtau,ss [ng*h/mL] | 1001002 | | xxxx | xxx# | xxx# | xxxx | XXX | XXX | XXX | XXX |
| Dose normalized AUCtau,ss, norm [ng*h/mL] | 1001002 | | | xxx | xxx | | xxx | xxx | xxx | xxx |
| tmax,ss [h] | 1001002 | | XXXX | XXX | XXX | xxx | XXX | XXX | | |

# = Obtained from implausible plasma concentration
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Programming note: List by parameter, then by subject. Do not display ratios for t\_max.

Statistical Analysis Plan Doc No D-18.239

### L PK RATIO

ACT-293987 Protocol: AC-065A309 Listing of Cmax,ss and AUCtau,ss ratio of ACT-333679/selexipag

Analysis Set: Pharmacokinetic Analysis Set

| | | | max,ss Ratio<br>33679/selexipag | AUCtau,ss Ratio<br>ACT-333679/selexipag | |
|---|---|---|---|---|---|
| Dose [ug bid] | Subject number | Uptravi | i.v. selexipag | Uptravi | i.v. selexipag |
| 200 ug b.i.d. p.o. / 225 ug b.i.d. i.v. | 1001002<br>1001003 | XXX<br>XXX | xxx<br>xxx | xxx#<br>xxx | xxx<br>xxx |
| | 1001005 | XXX | XXX | XXX | XXX |
| 400 ug b.i.d. p.o. / 450 ug b.i.d. i.v. | 1001004<br>1001010 | xxx<br>xxx | xxx<br>xxx | XXX | XXX<br>XXX |
| | 1001006 | XXX | xxx | XXX | xxx |
| Dose Normalized | 1001002<br>1001003<br>1001004<br>1001005 | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | xxx#<br>xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx<br>xxx |

# = Obtained from at least one impalusible plasma concentration
Output: <Output name>, Produced by DATAMAP on ddMMyyyy hh:mm (CET),
SDTM Date: ddMMyyyy
Program: /<folder>/program\_name>.sas
Page x of y

Programming note: List by dose, then by subject. Only list subjects who provided steady state data.

# $L_IMP_CONC$

ACT-293987

Protocol: AC-065A309

Listing of selexipag concentration in the infusion solution

Analysis Set: Pharmacokinetic Analysis Set

| Subject number | Visit / Time point | Selexipag concentration (eCRF) [ug] | Actual selexipag concentration [ug] |
|---|---|---|---|
| 1001002 | Visit 2 - Day 2 IV-1 | XXX | xxx |
| | Visit 2 - Day 2 IV-2 | XXX | XXX |
| | Visit 2 - Day 3 IV-3 | XXX | XXX |
| 1001003 | Visit 2 - Day 2 IV-1 | xxx | XXX |
| | Visit 2 - Day 2 IV-2 | XXX | XXX |
| | Visit 2 - Day 3 IV-3 | XXX | XXX |
| 1001006 | | | |

Actual selexipag concentration was assessed using a validated liquid chromatography with UV detector assay. Output: (Output name), Produced by DATAMAP on ddMMMyyyy hh:mm (CET), SDTM Date: ddMMMyyyy
Program: /<folder>//program\_name>.sas
Page x of y

Programming note: List by subject. Only list subjects who provided data. Layout may change slightly depending upon data structure.

# Appendix F Document history

Summarize the main changes and rationale for changes from one approved version to the next.

| Version | Effective Date | Reason |
|---|---|---|
| 1.0 | 22-May-2018 | New |
| | 2-Jul-2018 | Section 7.8.4: Implausible PK plasma concentrations will be identified by a PK specialist and flagged. PK parameters derived from implausible concentrations will be flagged as well. Flagged values will be listed but not included in summaries and statistical analyses. |
| | | Section 5.4.5.1: Added Uptravi in list of PAH-specific therapies to be displayed in the tables. |
| | | Section 8.2.2.4: Removed SAS code as this code will produce incorrect analysis (two-sample test / CI for median, while one-sample test / CI is appropriate). |
| 2.0 | | Section 8.2.3.3: Added j subscript for random intercept parameter for clarification of random parameter. |
| | | Section 12.4.1: Added clarification that tables will be run on the SAF and only on the ivSAF if different from SAF to be consistent with Table 4. |
| | | T_PK_EP_SUM: Removed ratio and CVb(%), as this information is contained in T_CV_MM. |
| | | Listings L_EG, L_EG_QUAL, L_MH: General medical history and ECG are not collected for screen failures, thus population is changed from SCR to SAF. |
| | | Corrections and additions to table shells to improve readability (e.g., date/time columns added, footnotes added) |